## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A multicentre, randomised, double-blind (sponsor-unblinded), placebo-controlled study to investigate the safety and tolerability, pharmacokinetics, pharmacodynamics, and efficacy of GSK2982772 in subjects with moderate to severe rheumatoid arthritis. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2982772 |
| <b>Effective Date</b> | : | 17-DEC-2018 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2015N251670\_03 and 2015 2015N251670\_04 in Germany.
- This RAP is intended to describe the safety, tolerability, PK, PD, and efficacy analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## Author(s)

| Author | |
|-----------|----------------------------------------|
| Lead | PPD |
| | Statistics Leader (Biostatistics) |
| Co-author | PPD |
| | Principal Statistician (Biostatistics) |

# RAP Team Review Confirmation (Method: E-mail)

| Reviewer | | Date |
|---|---|---|
| PPD | | 04- DEC-2018 |
| Principal Pro | Principal Programmer/Analyst (Clinical Programming) | |
| PPD | | 11- DEC-2018 |
| Director (CPI | MS) | 11- DEC-2016 |
| PPD | | 06-DEC-2018 |
| Clinical Deve | lopment Director (R&D Immuno-Inflammation) | 00-DEC-2016 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date | |
|-----------------|----------------------------------|-------------|
| Senior Statis | tics Director (Biostatistics) | 17-DEC-2018 |
| PPD Programming | g Manager (Clinical Programming) | 17-DEC-2018 |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | CLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | 2.2. | Study Objective(s) and Endpoint(s) Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| | ۷.4. | Statistical Hypotheses / Statistical Arialyses | 10 |
| 3. | | INED ANALYSES | 11 |
| | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | 11 |
| 4. | ANAL | YSIS POPULATIONS | 11 |
| •• | 4.1. | Protocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 40 |
| | 5.1. | VENTIONSStudy Treatment & Sub-group Display Descriptors | |
| | 5.1.<br>5.2. | Baseline Definitions | |
| | 5.2. | 5.2.1. Derivations and Handling of Missing Baseline Data | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | J. <del>4</del> . | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | 0.0. | Conventions | 15 |
| _ | OTUD | NV DODUH ATION ANALYOFO | 40 |
| 6. | | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | 16 |
| 7. | SAFE | TY ANALYSES | 16 |
| | 7.1. | Adverse Events Analyses | 16 |
| | 7.2. | Clinical Laboratory Analyses | |
| | 7.3. | Other Safety Analyses | |
| | 7.4. | Cardiovascular Events | 16 |
| 8. | EEEI | CACY ANALYSES | 17 |
| Ο. | 8.1. | | |
| | 0.1. | Efficacy Endpoints | |
| | | 8.1.1. Population of Interest | |
| | | 8.1.2.1. Statistical Methodology Specification | |
| | 8.2. | Exploratory Posterior Probabilities | |
| | · | | |
| 9. | PHAR | RMACOKINETIC ANALYSES | |
| | 9.1. | Primary Pharmacokinetic Analyses | |
| | | 9.1.1. Endpoint / Variables | |
| | | 9.1.1.1. Drug Concentration Measures | 20 |

## CONFIDENTIAL

203168

| | 9.2. | Population | n PK Analy | of Interestses | 20 |
|---|---|---|---|---|---|
| | 9.3. | PK/PD | | | 20 |
| 10 | DIOM | | IALVOEC | | 24 |
| 10. | 10.1. | | | | |
| | 10.1. | 10.1.1. | | Variables | |
| | | 10.1.1. | | of Interest | |
| | | 10.1.2. | | Analyses / Methods | |
| | | 10.1.5. | | Statistical Methodology Specification | |
| | 10.2. | Tarnet F | ngagement | Statistical Methodology Specification | 21 |
| | 10.2. | 10.2.1. | | Variables | |
| | | 10.2.2. | | of Interest | |
| | | 10.2.3. | | Analyses / Methods | |
| | | | | Statistical Methodology Specification | |
| | 10.3. | Transcrin | tomics Ana | lyses- mRNA from Blood | 24 |
| | | 10.3.1. | | Variables | |
| | | 10.3.2. | | of Interest | |
| | | 10.3.3. | | Analyses / Methods | |
| | | | | Fold Change Analysis | |
| | | | 10.3.3.2. | Microarray: Percentage inhibition | 27 |
| | | | | , | |
| 11. | REFE | RENCES. | | | 28 |
| 40 | 40051 | IDIOEO | | | - |
| 12. | | | | Desiries Management and Definition for Des | 29 |
| | 12.1. | Appendix | (1: Protocol | Deviation Management and Definitions for Per | 00 |
| | | | | from Day Dysterael Day Johns | |
| | 12.2 | | | from Per Protocol Population | |
| | 12.2. | Appendix | Drotocal Dr | le of Activitiesefined Schedule of Events | 3U |
| | 12.3. | | | ment Windows | |
| | 12.3. | | | of Assessment Windows for Analyses | |
| | 12.4. | | | hases and Treatment Emergent Adverse | 34 |
| | 12.4. | | | | 35 |
| | | 12.4.1. | | Ses | |
| | | 14.7.1. | | Study Phases for Concomitant Medication | |
| | | 12.4.2. | | Emergent Flag for Adverse Events | |
| | | | | States for AE Data | |
| | 12.5. | Appendix | | splay Standards & Handling Conventions | |
| | 12.0. | 12.5.1. | Reporting I | Process | 36 |
| | | 12.5.2. | | Standards | |
| | | 12.5.3. | | Standards for Pharmacokinetic | |
| | 12.6. | | | and Transformed Data | |
| | | 12.6.1. | | | |
| | | 12.6.2. | Study Popu | ulation | 39 |
| | | 12.6.3. | | | |
| | | | | HAQ-DI | |
| | | | 12.6.3.2. | Patient Global Assessment | 42 |
| | | | | Physician Global Assessment (PGA) | |
| | | | | Disease Activity Score (DAS28): | |
| | | | 12.6.3.5. | ACR Response Rates | 43 |
| | | | 12.6.3.6. | Swollen and Tender/Painful Joint Count | 44 |

## CONFIDENTIAL

| 00 | 2 | 168 |
|----|-----|-----|
| 71 | 1.5 | ınz |

| | | 12.6.3.7. | FACIT-Fatigue | 45 |
|---|---|---|---|---|
| | | 12.6.3.8. | | |
| | | 12.6.3.9. | CDAI and SDAI | 46 |
| | 12.6.4. | Safety | | 46 |
| | 12.6.5. | Biomarker | | 47 |
| | 12.6.6. | | | |
| 12.7. | Appendix | 7: Reporti | ng Standards for Missing Data | 49 |
| | 12.7.1. | Premature | : Withdrawals | 49 |
| | 12.7.2. | | of Missing Data | |
| | | 12.7.2.1. | Handling of Missing and Partial Dates | 49 |
| 12.8. | Appendix | 8: Values | of Potential Clinical Importance | <mark>5</mark> 0 |
| | 12.8.1. | | / Values | |
| | 12.8.2. | | | |
| | | | 3 | |
| 12.9. | | | viations & Trade Marks | |
| | 12.9.1. | | ons | |
| | 12.9.2. | | (S | |
| 12.10. | | | Data Displays | |
| | | | ay Numbering | |
| | | | mple Shell Referencing | |
| | | | es | |
| | | | ulation Tables | |
| | | | ables | |
| | | • | gures | |
| | | | oles | |
| | | | ures | |
| | | | kinetic Tables | |
| | | | kinetic Figures | |
| | | | kinetic/Pharmacodynamic Figures | |
| | | | Tables | |
| | 12.10.13 | .Biomarker | Figures | <mark>77</mark> |
| | | | gs | |
| | | | istings | |
| 12.11. | Appendix | : 13: Exam | ole Mock Shells for Data Displays | 86 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology | Revision Chronology: | |
|---|---|---|
| 2015N251670_00 | 01-APR-2016 | Original |
| 2015N251670_01 | 25-MAY-2016 | Protocol Amendment 1 incorporates the addition of risk text for drug interaction with Pglycoprotein (Pgp) inhibitors and narrow therapeutic index (NTI) CYP3A4 substrates, an updated list of prohibited medications plus some minor protocol clarifications and administrative changes. |
| 2015N251670_02 | 14-JUL-2016 | Protocol Amendment 02 incorporates the addition of suicidal ideation and behaviour (SIB) withdrawal criteria plus other minor protocol clarifications and administrative changes. |
| 2015N251670_03 | 20-APR-2017 | Protocol Amendment 03 incorporates the change in dosing regimen from 60 mg BID to 60 mg TID, restrictions on JAK inhibitors, defined non-reproductive potential criteria in Exclusion 11, change to clinical laboratory criteria in Exclusion 23, change in Haematologic Stopping Criteria in Section 5.4.5, addition of evaluation of joint space narrowing with MRI, flexibility in scheduling with MRI and synovial biopsy, some minor protocol clarifications and administrative changes. |
| 2015N251670_04 | 03-AUG-2017 | Protocol Amendment 04 incorporates a country specific amendment for Germany which reinstates the clinical laboratory criteria in Exclusion 23 and Haematologic Stopping Criteria in Section 5.4.5 that was changed in Amendment 03. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| A formal interim analysis will<br>be conducted during the study.<br>The timing of this analysis will<br>either be on the<br>recommendation of the data<br>review group to assess futility | A formal interim analysis will no longer be conducted based on review of recruitment information and recommendation by the DRC | Quick recruitment towards the end of the study meant that timelines for the interim analysis would occur after all subjects had completed the treatment phase of the study, therefore leaving no ability to stop the |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| based on 6 weeks of treatment, or when an appropriate number have completed 12 weeks of treatment, whichever is earliest. The purpose of the Interim Analysis would be to assess whether to stop the study for futility. This interim analysis may also facilitate decision making regarding the subsequent clinical development of GSK2982772 for RA. | | study for futility |
| Exploratory endpoint defined as change from baseline in RA symptom questionnaire score Exploratory endpoints: Inflammatory biomarkers, pathway engagement and mRNA in synovial tissue. | An overall score will not be provided due no available rules for how to combine these questions together, instead each item will be summarised separately These endpoints will not be analysed due to very small sample size and therefore lack of sufficient data to enable statistical analysis to be conducted. | Development of the questionnaire still in progress and no scoring system currently in place. Therefore no overall questionnaire score can be calculated. Uptake from subjects in the study to provide the optional synovial tissue samples was very limited. Only 5 subjects consented with only three of these providing a baseline and end of treatment sample. The decision therefore was made by the team not to perform the lab analysis of these samples, therefore planned analysis |
| | | cannot be conducted. Synovial tissue samples will still be used to explore PK concentration and Target engagement |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To investigate the safety and tolerability of 60 mg three times daily doses of GSK2982772 in subjects with moderate to severe Rheumatoid Arthritis. | <ul> <li>Adverse events.</li> <li>Clinical laboratory values (clinical chemistry, haematology and urinalysis).</li> <li>Vital sign measurements (blood pressure, heart rate, respiratory rate, and body temperature).</li> <li>12-Lead ECG monitoring.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To investigate the plasma concentrations of GSK2982772 following 60 mg three times daily doses of GSK2982772 in subjects with moderate to severe Rheumatoid Arthritis.</li> <li>To investigate the effect of 60 mg three times daily doses of GSK2982772 on inflammatory biomarkers in blood subjects with moderate to severe Rheumatoid Arthritis.</li> </ul> | <ul> <li>Pre-dose concentrations of GSK2982772 on Days 8, and 43 (Week 6).</li> <li>Post-dose concentrations of GSK2982772 on Days 1, 8, and 43 (Week 6) at 1, 2, 4 and 6 hours.</li> <li>Trough concentrations on Day 85 (Week 12).</li> <li>Change from baseline in blood inflammatory markers (e.g., may include but not limited to CRP, IL6, MMP-1, MMP-3, MMP-13, TIMP-1, MCP-1, MIF, MRP8/14 and other markers encompassed by Vectra DA).</li> </ul> |
| To investigate the effect of 60 mg three times daily doses of GSK2982772 on bone and synovial parameters as measured by MRI and DCE-MRI in subjects with moderate to severe Rheumatoid Arthritis. | Change from baseline in MRI parameters in the most affected hand/wrist. MRI parameters may include assessment of bone erosions, synovitis, bone oedema and joint space narrowing as assessed in the OMERACT-RAMRIS (Outcome Measures in Rheumatology, Rheumatoid Arthritis Magnetic Resonance Image Scoring System) scoring system, the RAMRIQ (rheumatoid arthritis MRI quantitative) scoring system, the modified CARLOS (Cartilage Loss Scoring System) and additional exploratory endpoints as data permit. |
| | <ul> <li>Change from baseline in synovial inflammation as measured by dynamic contrast enhanced (DCE)-MRI in the most affected hand/wrist:</li> <li>Exchange rate (K<sup>trans</sup>)</li> <li>Interstitial volume (V<sub>e</sub>)</li> <li>Plasma volume (V<sub>p</sub>)</li> <li>Initial rate of enhancement (IRE)</li> <li>Maximal signal intensity enhancement (ME)</li> <li>Joint volume</li> <li>Enhancing volume</li> </ul> |
| To investigate the effect of 60 mg<br>three times daily doses of<br>GSK2982772 on clinical disease<br>activity in subjects with moderate<br>to severe Rheumatoid Arthritis. | <ul> <li>Change from baseline in Disease Activity Score (DAS) 28-CRP scores.</li> <li>Proportion of subjects achieving categorical DAS28-CRP response (moderate/good EULAR response) at each assessment time points.</li> <li>Proportion of subjects achieving categorical</li> </ul> |
| To investigate the effect of 60 mg<br>three times daily dosing of<br>GSK2982772 on methotrexate<br>(MTX) concentrations | ACR20/50/70 response. Plasma concentrations of MTX pre-dose GSK2982772 on Days 1, 8, and 43 (Week 6). |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To investigate the effect of 60 mg three times daily doses of GSK2982772 on inflammatory biomarkers in synovial tissue in subjects with moderate to severe Rheumatoid Arthritis. | Change from baseline in CD68+ macrophages,<br>CD55+ fibroblast-like synoviocytes and a number of<br>infiltrating CD3, CD22, CD138 inflammatory cells,<br>and synovial inflammatory biomarkers including, but<br>not limited to VEGF, IL-1β, IL-6, TNFα, and MMP-1. |
| To investigate pathway and target<br>engagement following 60 mg three<br>times daily doses of GSK2982772<br>in blood and synovial tissue in<br>subjects with moderate to severe<br>Rheumatoid Arthritis. | <ul> <li>Pharmacology biomarker endpoints may include, but are not limited to the following, pre-dose at Days 1, 43 (Week 6) and trough on Day 85 (Week 12), as applicable and if evaluable samples and data permit:</li> <li>Target Engagement Assay RIP1 (TEAR1) in blood and synovial tissue.</li> </ul> |
| | Total or phosphorylated RIP1, MLKL, and RIP3, cleaved and total caspase 3 and caspase 8 signatures in synovial tissue. |
| To investigate the concentration of<br>GSK2982772 and possible drug-<br>related material, as well as specific<br>distribution within tissue if feasible,<br>in the synovial tissue after 60 mg<br>three times daily doses of<br>GSK2982772. | Pre-dose GSK2982772 synovial tissue biopsies and possible drug-related material concentrations, as well as specific distribution within tissue if feasible, on Day 43 (Week 6), as evaluable samples and data permit |
| To investigate the effect of 60 mg<br>three times daily doses of<br>GSK2982772 on the quality of life | Change from baseline in Health Assessment<br>Questionnaire Disability Index (HAQ-DI). |
| of subjects with moderate to severe Rheumatoid Arthritis. | Change from baseline in RA symptom questionnaire score. |
| | Change from baseline in Functional Assessment of<br>Chronic Illness Therapy (FACIT)-Fatigue. |
| To investigate the effect of 60 mg three times daily doses of GSK2982772 on gene expression in the blood of subjects with moderate to severe Rheumatoid Arthritis. | Transcriptomic analysis of mRNA isolated<br>from blood pre-dose on Days 1 and 43<br>(Week 6) and trough on Day 85 (Week 12). |
| To investigate the effect of 60 mg three times daily doses of GSK2982772 on gene expression in synovium of subjects with moderate to severe Rheumatoid Arthritis. | • Transcriptomic analysis of mRNA isolated from synovial tissue pre-dose on Days 1 and 43 (Week 6). |

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

The primary objective of the study is to investigate the safety and tolerability of GSK2982772 following 12 weeks of treatment. No formal statistical hypotheses will be conducted to assess this objective.

If appropriate, comparisons between the GSK2982772 and the placebo arm will be made to investigate the secondary pharmacodynamic, mechanistic and efficacy objectives. Trends over time will be investigated for both treatment arms along with associations between each of the pharmacodynamic, mechanistic and efficacy parameters.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal interim analysis will be conducted. Details of decision to not conduct the planned interim analysis provided in Section 2.1.

Unblinded biomarker, efficacy and pharmacodynamic analyses will be conducted and delivered to the data review committee (DRC) according to the DRC charter. Safety will also be evaluated in the context of the pharmacodynamic, biomarkers and efficacy observed.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | Comprises of all subjects who were screened for the study | Selected Accountability data |
| Randomised | Comprises of all subjects who were randomised | All listings unless specified |
| Safety | <ul> <li>Comprise of all subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject was randomised to.</li> </ul> | <ul><li>Demography</li><li>Safety</li><li>Efficacy</li><li>Exploratory</li><li>Biomarker</li></ul> |
| Pharmacokinetic<br>GSK298772<br>(PK772) | Subjects in the 'Safety' population who received<br>an active dose and for whom a GSK2982772<br>pharmacokinetic sample was obtained and<br>analysed. | • GSK2982772 PK |
| Pharmacokinetic<br>Methotrexate<br>(PKMeth) | Subjects in the 'Safety' population who received<br>an active dose and for whom a Methotrexate<br>pharmacokinetic sample was obtained and<br>analysed. | Methotrexate PK |
| Per-Protocol (PP) | Subjects in the 'Safety' population with those who had an important deviation with potential to | DAS28-CRP |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | impact the analysis excluded. Please see Section 12.1.1 for definition of deviations that lead to | |
| | exclusion from this population. | |
| PP completers | All subjects in the PP population who also complete the study. [1] | DAS28-CRP |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

[1] Completion of the study as defined from the eCRF study conclusion page.

Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK Display Standards and CDISC SDTM/ADaM standards

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [02OCT18 and Version 3].

- Data will be reviewed prior to freezing the database to ensure all important are captured and categorised on the protocol deviations dataset. This dataset will also be reviewed to ensure exclusions from any populations are documented appropriately.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | | | |
|---|---|---|---|---|---|
| [RandAl | I NG / FSO Randomization<br>System] | Data Displays for Reporting | | | |
| Code | Description | Description Description in tables/figures (TRTGRP) Order in | | Description in Listings<br>(ATRTGRP) | Order<br>in<br>Outputs |
| А | GSK2982772 BID 60<br>mg | GSK2982772 60mg | 2 | GSK2982772 60mg<br>BID | 3 |
| С | GSK2982772 60mg<br>TID | GSK2982772 60mg | 2 | GSK2982772 60mg<br>TID | 4 |
| Р | Placebo | Placebo | 1 | Placebo BID | 1 |
| Q | Placebo TID | Placebo | 1 | Placebo TID | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

## 1. GSK2982772 60mg vs Placebo

If a subject is found to have received incorrect medication at all during their study duration all of their data will be analysed/summarised according to the treatment group, they were randomised to. A listing of planned and actual treatments will be provided identifying any subjects who did indeed receive incorrect medication.

A couple of the key efficacy endpoints will be summarised separately for the BID and TID treatment regimens, details are provided in Appendix 12: List of Data Displays.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Assessme<br>Ba | Baseline Used in<br>Data Display | |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Safety | | | |
| Vital Signs <sup>[1,2]</sup> | Х | Х | Day 1 (Pre-Dose) |
| 12-Lead ECG <sup>[2]</sup> | X[3] | Х | Day 1 (Pre-Dose) |
| Clinical Laboratory<br>Values <sup>[2,4]</sup> | Х | X | Day 1 (Pre-Dose) |
| Columbia Suicide<br>Severity Rating Scale (C-SSRS) | Х | Х | Day 1 (Pre-Dose) |

| Parameter | Study Assessme<br>Ba | Baseline Used in<br>Data Display | |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | _ |
| Secondary | | · | |
| Plasma concentrations of GSK2982772/MTX | | X | Day 1 (Pre-Dose) |
| Inflammatory Biomarkers in Blood | | X | Day 1 (Pre-Dose) |
| MRI/DCE-MRI | | X | Day 1 (Pre-Dose) |
| DAS28(CRP) | | Х | Day 1 (Pre-Dose) |
| ACR20/50/70 | | Х | Day 1 (Pre-Dose) |
| Exploratory | | | |
| Pharmacology<br>Biomarkers in Blood | | X | Day 1 (Pre-Dose) |
| Concentration of<br>GSK2982772 and<br>Possible Drug-Related<br>Material in the Synovial<br>Tissue | | X | Day 1 (Pre-Dose) |
| HAQ-DI | | X | Day 1 (Pre-Dose) |
| RA Symptom<br>Questionnaire | | X | Day 1 (Pre-Dose) |
| (FACIT)-Fatigue | | X | Day 1 (Pre-Dose) |
| Physician Global<br>Assessment | | X | Day 1 (Pre-Dose) |
| Patient Global<br>Assessment | | X | Day 1 (Pre-Dose) |
| mRNA in Blood | | X | Day 1 (Pre-Dose) |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- [1] Vital sign measurements include Blood Pressure, Heart Rate, Respiratory Rate, and Body Temperature.
- [2] Where both screening and pre-dose are available, the value closest to first dose will be used.
- [3] ECG recordings will be performed in triplicate at screening. Use the mean of the triplicate measurements.
- [4] Clinical Laboratory measurements include Clinical Chemistry, Haematology and Urinalysis.
- For Safety Data, If Day 1 pre-dose is missing then Screening will be used as baseline
- For Safety Data, If Day 1 is Post Dose, Screening will be used as baseline

### 5.2.1. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

## 5.3. Multicentre Studies

There are no planned adjustments for multiple centres or regions due to the size of the study. For all analyses all sites, countries and regions will be pooled.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

| Category | Details |
|------------|--------------------------------------------------|
| Strata | Not applicable for this study |
| Covariates | Baseline measure will be included as a covariate |

## 5.4.2. Examination of Subgroups

There are no planned subgroup analyses to be conducted on this study.

## 5.5. Multiple Comparisons and Multiplicity

Unless specified no adjustments will be made for multiple comparisons or multiplicity.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK Display Standards and CDISC SDTM/ADaM standards

## 7. SAFETY ANALYSES

The safety analyses will be based on the safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse event analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 7.4. Cardiovascular Events

If any of the following events are recorded in the eCRF as a CV event during the study further patient profiles will be generated according to IDSL and provided to the GCSP department: Arrhythmias, Congestive heart failure, Cerebrovascular events/stroke and Transient ischemic attack (TIA), Deep vein thrombosis (DVT)/Pulmonary embolism (PE), Myocardial Infarction/Unstable Angina, Peripheral arterial thromboembolism, Pulmonary Hypertension, Revascularisation, Valvulopathy.

## 8. EFFICACY ANALYSES

# 8.1. Efficacy Endpoints

Table 2 Overview of Planned Efficacy Analyses

| Endpoint | Absolute | | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | Summary Individual | | Stats Analysis | | | Summary | | Individual | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Efficacy | | | | | | | | | | | | | | |
| FACIT-Fatigue | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| HAQ-DI | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| Patient Global | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| assessment | | | | ' | | | ' | ' | ' | ľ | ' | | | |
| Physician Global | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| Assessment | | | | Ī | | | _ | - | | | - | | | |
| DAS28-CRP | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| DAS28-CRP EULAR | | | | | | | | | | | Υ | | | Υ |
| response | | | | | | | | | | | | | | - |
| ACR Response Rates | | | | | | | | | | | Υ | | | Υ |
| TJC28 | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| SJC28 | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| MRI parameters <sup>2</sup> in most affected wrist | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| DCE-MRI <sup>3</sup> | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| Patient assessment of joint Pain | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| RA symptom questionnaire | | | | Υ | | | Υ | | | | | | | |
| CRP | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| CDAI <sup>4</sup> | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |
| SDAI <sup>4</sup> | | | | Υ | | | Υ | Υ | Υ | Υ | Υ | | | |

#### 1. NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- 2: Bone erosions, synovitis, bone oedema, joint space narrowing (Based on RAMRIS/RAMRIQ and CARLOS)
- 3: Exchange rate, Interstitial volume, plasma volume, initial rate of enhancement, maximal signal intensity enhancement, joint volume, enhancing volume
- 4: Although not listed in the protocol as endpoints, these were added to aide decision making at the administrative review and the end of the study.

## 8.1.1. Population of Interest

The efficacy analyses will be based on the safety population, unless otherwise specified.

## 8.1.2. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.1.2.1. Statistical Methodology Specification

#### Statistical Analyses (cts endpoints with mmrm analysis)

#### Secondary/exploratory Endpoint(s)

- Change from baseline (pre-dose Day 1) in FACIT-Fatigue score at Days 43 (pre-dose), and 85.
- Change from baseline (pre-dose Day 1) in HAQ-DI at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in Patient Global Assessment at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in Physician Global Assessment at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in DAS28-CRP at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in TJC28 at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in SJC28 at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in MRI parameters based on RAMRIS at days 43 (pre-dose) and 85.
- Change from baseline (pre-dose Day 1) in MRI parameters based on RAMRIQ at days 43 (pre-dose) and 85.
- Change from baseline (pre-dose Day 1) in MRI parameters based on CARLOS at days 43 (pre-dose) and 85.
- Change from baseline (pre-dose Day 1) in MRI parameters based on DCE-MRI at days 43 (pre-dose) and 85.
- Change from baseline (pre-dose Day 1) in patient assessment of pain at days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in CRP on days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in CDAI on days 15, 29, 43 (pre-dose), 57, 71, 85.
- Change from baseline (pre-dose Day 1) in SDAI on days 15, 29, 43 (pre-dose), 57, 71, 85.

#### **Model Specification**

- Endpoints will be statistically analyzed using a mixed models repeated measures (MMRM) approach.
- Terms fitted in the MMRM model will include:
  - Fixed Category : Treatment, Day, Treatment\*Day

Fixed Continuous Covariates : Baseline Score, baseline\*Day

Repeated Effect : Day

 The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

 An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line with a subject=SUBJID option.

Note: Other covariates maybe explored, if deemed appropriate for sensitivity analyses.

#### **Model Checking & Diagnostics**

- For the MMRM, model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- In the unlikely circumstance that there are convergence problems with the MMRM analysis, this will be explored. For example the SCORING=4 option could be used in the MIXED statement, which makes SAS use Fisher scoring for the first 4 iterations. If the convergence problem cannot be resolved, the unstructured covariance matrix will be replaced by ANTE(1) covariance structure in combination with a random subject effect.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.

Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- LS means and corresponding standard error of means (SEs) and 95% confidence intervals
  will be presented for each treatment by time interaction, together with estimated treatment
  differences (GSK2982772 Placebo) and the corresponding 95% confidence intervals will be
  produced.
- Observed Margins will be specified to produce the LS means.
- Plots of LS means and standard errors from the model will be generated over time by treatment.

## 8.2. Exploratory Posterior Probabilities

Decision criteria for this study will be based on posterior probabilities of treatment differences (GSK2982772 vs Placebo) for the following endpoints; DAS28 (CRP), ACR20 and ACR50. Posterior probabilities will explore the likelihood that the treatment difference is greater than X based on the data observed.

A Bayesian approach will be employed to determine a 95% credible confidence interval and the posterior probabilities assuming a noninformative prior: Beta (1, 1) for ACR analyses and N [0, 1.E36).for the analysis of the DAS28-CRP. Any such analyses will be done by GSK II Clinical Statistics for both the administrative review and SAC.

## 9. PHARMACOKINETIC ANALYSES

## 9.1. Primary Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

## 9.1.1.1. Drug Concentration Measures

Plasma Concentration data for GSK2982772 will be summarised and listed, no statistical analysis will be conducted. Summary statistics of GSK2982772 concentration by Day (1, 8, 43 and 85) and nominal blood sampling time (pre-dose, and 1, 2, 4 and 6 hours post-dose) will be determined.

Plasma concentration data for methotrexate will be summarised and listed, no statistical analysis will be conducted. Summary statistics of methotrexate pre-dose concentrations by Day (1, 8 and 43) will be determined.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic).

#### 9.1.2. Population of Interest

All PK statistical displays will be based on the ["PK772"] population, unless otherwise specified.

## 9.2. Population PK Analyses

GSK2982772 plasma concentrations from this study may be included in a cross-study population pharmacokinetic analysis after SAC. To support this analysis a NONMEM datafile will be generated. The details for the dataset specifications will be provided by CPMS after SAC, if needed.

#### 9.3. PK/PD

Concentration data and blood/synovial fluid target engagement will be explored graphically.

Concentration data will also be presented graphically against change from baseline in DAS28 (CRP) by visit.

#### 10. BIOMARKER ANALYSES

#### 10.1. Biomarker

## 10.1.1. Endpoint / Variables

#### **Overview of Planned Biomarker Analyses**

| Endpoint | | Absolute | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | mary | mary Individual | | Stats Analysis | | | Summary | | Indiv | idual |
| | Т | T F L | | F | F | L | Т | T F L | | Т | F | F | L |
| <b>Secondary Biomarkers</b> | | | | | | | | | | | | | |
| Inflammatory biomarkers in blood <sup>1</sup> | | | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | | | |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
  - 1: Markers including CRP, CHI3L1, EGF, IL6, Leptin, MCP-1, MIF, MMP-1, MMP-3, MMP-13, Resistin, SAA, S100A8/S100A9, TIMP-1, TNF-RI, VCAM-1, VEGFA and unadjusted Vectra DA

## 10.1.2. Population of Interest

The biomarker analyses will be based on the "Safety" population, unless otherwise specified.

## 10.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1.will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 10.1.3.1. Statistical Methodology Specification

#### **Inflammatory Blood Biomarkers**

#### Endpoint(s)

Change from baseline on log transformed inflammatory biomarkers in blood on Day 43 and 85 pre-dose: Loge Change = Loge (Visit) – loge (Baseline)

1. Markers: CRP, CHI3L1, EGF, IL6, Leptin, MCP-1, MIF, MMP-1, MMP-3, MMP-13, Resistin, SAA, S100A8/S100A9, TIMP-1, TNF-RI, VCAM-1, VEGFA and unadjusted Vectra DA

## **Model Specification**

 Endpoints will be statistically analyzed using a mixed models repeated measures (MMRM) approach. Terms fitted in the MMRM model will include:

Fixed Category : Treatment, Day, Treatment\*Day
 Fixed Continuous Covariates : Baseline Score, baseline\*Day

Repeated Effect : Day

 The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

 An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line with a subject=SUBJID option.

#### **Model Checking & Diagnostics**

- For the MMRM, model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- In the unlikely circumstance that there are convergence problems with the MMRM analysis, this will be explored. For example, the SCORING=4 option could be used in the MIXED statement, which makes SAS use Fisher scoring for the first 4 iterations. If the convergence problem cannot be resolved, the unstructured covariance matrix will be replaced by ANTE(1) covariance structure in combination with a random subject effect.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.

Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### Presentation of results

- Adjusted geometric means for each treatment group at each timepoint and associated 95% confidence interval will be constructed by back transforming the LS means from the model.
- ➤ The treatment ratios and 95% CI will be calculated by back-transforming the difference in the LS means (GSK2982772 Placebo) and associated 95% CI

Percentage change from baseline at each timepoint will be calculated using the formula: 100% x (exp(LS mean)- 1)

Plots of LS means and standard errors from the model will be generated over time by treatment.

## 10.2. Target Engagement

### 10.2.1. Endpoint / Variables

#### Table 3 Overview of Planned Target Analyses

| Endpoint | | Absolute | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | Summary Individual | | ridual | Stats Analysis | | | Summary | | Indiv | idual |
| | Τ | F | L | Т | F | F | L | Τ | F | L | Т | F | F | L |
| Target Engagement | | | | | | | | | | | | | | |
| target engagement in blood <sup>3</sup> | | | | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | | | |
| target engagement in synovial tissue <sup>3</sup> | | | | | | | Υ | | | | | | | |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- 3: TEAR1 in blood and synovial tissue, Free RIP1 and Total RIP1.
   1.

## 10.2.2. Population of Interest

The target/pathway engagement analyses will be based on the "Safety" population, unless otherwise specified.

## 10.2.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 10.2.3.1. Statistical Methodology Specification

## **Target Engagement**

#### **Endpoints**

Log Ratio = Log (free TEAR1) – log (total TEAR1)

.

#### **Model Specification**

- A mixed effect model will be fitted with treatment, time (i.e. planned relative time) and treatment \* time as a fixed effect and subject as a random effect. Baseline log ratio will be fitted as a continuous covariate along with Baseline log ratio\* time.
- > The Kenward and Roger method for approximating the denominator degrees of freedom and

### **Target Engagement**

correcting for bias in the estimated variance-covariance of the fixed effects will be used.

An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line with a subject=SUBJID option.

#### **Model Checking**

- For the MMRM, model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- In the unlikely circumstance that there are convergence problems with the MMRM analysis, this will be explored. For example, the SCORING=4 option could be used in the MIXED statement, which makes SAS use Fisher scoring for the first 4 iterations. If the convergence problem cannot be resolved, the unstructured covariance matrix will be replaced by ANTE(1) covariance structure in combination with a random subject effect.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.

Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

➤ If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Presentation of Results**

- Engagement ratio relative to baseline and associated 95% confidence interval will be calculated for each post-baseline timepoint, using the formula exp(ln(ratiopost/ratiopaseline) +1).
- Percentage target engagement at each timepoint will be calculated from the adjusted geometric means using the formula (1-engagment ratio)\*100%.
- ➤ The treatment engagement ratios and 95% CI will be calculated by back-transforming the difference between the least square means and associated 95% CI
- The treatment difference percentage target engagement is (1 treatment engagement ratio) \* 100%

## 10.3. Transcriptomics Analyses- mRNA from Blood

RNA will be extracted and hybridised using a balanced batch design by Epistem. Microarray mRNA data will be normalised using gcRMA or RMA in Array Studio v5.0 or later. After normalisation, the data will be quality assessed and any samples deemed as QC fails will be excluded from any further analysis. This quality assessment will involve looking for outlying signals in both the normalised expression data and the MAS5 QC metrics generated from each sample. If any samples are excluded, the remaining data will be re-normalised. The output from the normalisation will be log<sub>2</sub> transformed mRNA intensity data (measured in arbitrary units).

Microarray data consists of expression values (log<sub>2</sub>-transformed) derived from individual probesets designed against coding regions of individual genes. More than one probeset

can exist per gene. This analysis will be conducted at the probeset level. The probeset, gene or gene description will be included in the outputs.

In order to identify the most robustly expressed probesets, the data can be filtered to remove low intensity probesets, low quality and control probe sets prior to analysis. This could be done simply by excluding all probesets where all observations are <6 (on the log<sub>2</sub> scale). Note it has been observed empirically that when you get below 100 (6.6 on the log<sub>2</sub> scale) you are into the noise of the assay. Other more stringent methods of filtering the data could be used. In total there are 53,617 probesets that could be analysed.

mRNA data is available from blood samples only as described in Section 2.1. mRNA summaries and listings will be the responsibility of the GSK stats and programming team and will be delivered at an agreed date after SAC.

## 10.3.1. Endpoint / Variables

### **Overview of Planned Biomarker Analyses**

| Endpoint | | | A | Absolu | ite | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | | mary | y Individual Stats Analys | | lysis | Sum | mary | Individua | | | |
| | Τ | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Transcriptomics | | | | | | | | | | | | | | |
| mRNA from blood <sup>4</sup> | | | | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | | | |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- 4: Data to be provided by Epistem and analysed by the GSK stats and programming team
   1.

## 10.3.2. Population of Interest

The transcriptomic analyses will be based on the "Safety" population, unless otherwise specified.

#### 10.3.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. Note that probeset ID is required to be included in analyses and outputs if there is more than one probeset per gene.

### **Primary Statistical Analyses**

#### Endpoint(s)

- Log2(intensity) mRNA expression of inflammatory gene transcripts
- Percentage inhibition of inflammatory gene transcripts

## **Model Specification**

- Endpoints will be statistically analyzed using a linear repeated measures mixed effects model.
- Terms fitted in the linear repeated measures mixed effects model will include:

Fixed Category : Treatment, Visit, Treatment \* Visit

Random Effect : Subject

## **Model Checking & Diagnostics**

- For the MMRM, model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- In the unlikely circumstance that there are convergence problems with the MMRM analysis, this will be explored. For example, the SCORING=4 option could be used in the MIXED statement, which makes SAS use Fisher scoring for the first 4 iterations. If the convergence problem cannot be resolved, the unstructured covariance matrix will be replaced by ANTE(1) covariance structure in combination with a random subject effect.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.

Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

➤ If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Presentation of Results**

- For each probeset analysed, adjusted means with corresponding 95% CI and fold changes (for Log2(intensity)) or difference in LS means (for Percentage inhibition) with corresponding 95% CI's can be outputted. The fold change is derived from the ratio of the back-transformed estimate of the difference between LS means.
- Plots of LS means and standard errors from the model will be generated for each treatment by time.

#### 10.3.3.1. Fold Change Analysis

The log<sub>2</sub> normalised copy numbers (also referred to as log2(intensity)) received from the normalised process will be listed and summarised appropriately.

As the data will be  $\log_2$  transformed prior to the analysis the treatment effects will be expressed as ratios after back transformation to the original scale. These ratios can be converted from treatment ratios to fold change values as follows:

- If ratio  $\geq 1$  then fold change = ratio
- If ratio < 1 then fold change = -1/ratio

To compare the expression value for each probeset, the following linear repeated measures mixed effects model will be fitted to each probeset that passes any pre-filtering, with log2 (intensity) as the response variable as outlined in Section 10.3.3. Where appropriate, particularly with microarray data, multiple testing will be taken into account using the Benjamini-Hochberg correction [Benjamini, 1995] to calculate FDR adjusted p-values. A summary may be generated, including probeset ID, gene ID, time point, adjusted means with corresponding 95% CI for each treatment group, Benjamini-Hochberg FDR adjusted p-value and fold changes corresponding 95% CI from each comparison for probesets found to be significant after the applying the Benjamini-Hochberg correction.

For each comparison, subsets of probesets will be identified based on an appropriate fold-change, for example, fold changes >1.5 or <-1.5. The proportion of probesets with fold changes >1.5 or <-1.5 will be summarised in a frequency table.

Exploratory graphical reporting on the back-transformed scale can include:

- Log<sub>2</sub> (intensity) plotted against time point separately for individual subjects, grouped by treatment group
- Adjusted mean intensity and 95 CI% plotted by treatment group and time point

#### 10.3.3.2. Microarray: Percentage inhibition

Based on results from the fold change analyses, the selected probesets will be further explored through percentage inhibition. The log<sub>2</sub> normalised data is back transformed and the percentage inhibition is derived on a subject level on the back transformed data for each probeset. The percentage inhibition will be determined for each probeset per subject, where it is defined as the reduction from baseline. For example:

Day X – baseline = -40% would be a 40% reduction (i.e. -40% change from baseline) which in turn is defined as a 40% inhibition.

So the percentage inhibition would be calculated as:

[ (Day x – Baseline) / Baseline ] \* 
$$-100 = \%$$
 inhibition

A subset of probesets may be identified and individual subject mRNA intensities and percentage inhibitions may be listed, summarised and plotted appropriately for each selected probeset. The selected probesets will be statistically analysed appropriately, and the output from the mixed effects model (outlined in Section 10.3.3) summarised.

## 11. REFERENCES

Benjamini Y and Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. J Royal Stat Soc 1995;57:289-300

## 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 12.1.1. Exclusions from Per Protocol Population

Criteria for exclusion from the per protocol population are detailed in the protocol deviation management plan (PDMP). The stats and programming team will use the information in the protocol deviations dataset to select subjects who have deviations that are flagged as important and that should be removed from the per protocol population.

# 12.2. Appendix 2: Schedule of Activities

## 12.2.1. Protocol Defined Schedule of Events

| | 30) | | | | | | Trea | itment Po | eriod <sup>17</sup> | 7 | | | | | wal <sup>18</sup> | 3)19 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening (-30) | Day 1 | Day 8 (±3) | Day 15 (±3) | Day 22 (±3) | Day 29 (±3) | Day 36 (±3) | <b>Day 43 (±3)</b><br>(week 6) | Day 50 (±3) | Day 57 (±3) | Day 64 (±3) | Day 71 (±3) | Day 78 (±3) | <b>Day 85 (+2)</b> (week 12) | Early Withdrawal <sup>18</sup> | Follow Up (±3)¹9 |
| Site Visit | Χ | Χ | Χ | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | Χ | Х |
| Phone call | | | | | Χ | | Χ | | Χ | | Χ | | Χ | | | |
| General/Safety A | \sse | essme | nts a | and | Proc | edure | es | | | | | | | | | |
| Informed<br>Consent | Χ | | | | | | | | | | | | | | | |
| Subject<br>Demography | Х | | | | | | | | | | | | | | | |
| Full medical history <sup>1</sup> | Х | | | | | | | | | | | | | | | |
| Inclusion/Exclusi on Criteria | Х | | | | | | | | | | | | | | | |
| Full physical exam <sup>2</sup> | Х | | | | | | | | | | | | | Х | Χ | Χ |
| Brief physical exam | | X <sup>4</sup> | | Χ | | Χ | | X <sup>4</sup> | | Х | | Χ | | | | |
| Vital signs (BP,<br>HR, RR,<br>temperature) | Х | X <sup>4</sup> | Х | Х | | Х | | X <sup>4</sup> | | Х | | Х | | Х | Х | Х |
| 12-lead ECG | $X^3$ | $X^4$ | Χ | Χ | | Χ | | X <sup>4</sup> | | X | | Χ | | Χ | Χ | Χ |
| Concomitant<br>medication<br>review & AE<br>reporting/SAEs <sup>5</sup> | X | | | | | | | | X | | | | | | | |
| PROs/Questionr | naire | es/Dia | ries/ | Dise | ase | Asse | ssmen | ts and P | roced | ures | | | | | | |
| Columbia<br>Suicide Severity<br>Rating Scale (C-<br>SSRS) | Х | X <sup>4</sup> | | | | | | X <sup>4</sup> | | | | | | Х | Х | |
| FACIT-fatigue;<br>RA Symptom<br>and Impact<br>Diary <sup>6</sup> | | X <sup>4</sup> | | | | | | X <sup>4</sup> | | | | | | Х | X | |
| HAQ-DI; Patient<br>Assessment of<br>joint pain <sup>6</sup> | | X <sup>4</sup> | | Χ | | Х | | X <sup>4</sup> | | Χ | | Χ | | Χ | X | |
| Patient Global<br>Assessment<br>(PtGA) <sup>6</sup> | Χ | X <sup>4</sup> | | X | | Х | | X <sup>4</sup> | | Х | | Χ | | Х | Х | |

| | 30) | | | | | | Trea | tment P | eriod <sup>17</sup> | 7 | | | | | wal <sup>18</sup> | 3)19 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening (-30) | Day 1 | Day 8 (±3) | Day 15 (±3) | Day 22 (±3) | Day 29 (±3) | Day 36 (±3) | <b>Day 43 (±3)</b><br>(week 6) | Day 50 (±3) | Day 57 (±3) | Day 64 (±3) | Day 71 (±3) | Day 78 (±3) | <b>Day 85 (+2)</b> (week 12) | Early Withdrawal <sup>18</sup> | Follow Up (±3)¹ <sup>9</sup> |
| Tender (28) &<br>Swollen (28)<br>joint count | Х | X <sup>4</sup> | | Χ | | Х | | X <sup>4</sup> | | Х | | Х | | X | X | |
| Physician Global<br>Assessment<br>(PGA) | | X <sup>4</sup> | | Χ | | Х | | X <sup>4</sup> | | X | | Х | | Χ | Х | |
| MRI/DCE-MRI <sup>7</sup> | | X <sup>4</sup> ,<br>20 | | | | | | X <sup>4,21</sup> | | | | | | X <sup>22</sup> | X <sup>16</sup> | |
| Study Treatmen | t | | | | | | | | | | | | | | | |
| Randomisation | | Χ | | | | | | | | | | | | | | |
| Study<br>medication<br>(three times<br>daily) <sup>8</sup> | | X | | | | | | X | <br>( | | | | | | | |
| Dispensing of study medication | | Χ | | | | Χ | | | | Χ | | | | | | |
| Dispensing of diary cards | | Х | Χ | Χ | | X | | Х | | X | | Χ | | | | |
| Collection and review of diary cards | | | Χ | Χ | | Х | | Χ | | Χ | | Х | | X | X | |
| Laboratory (Safe | ety) | Asses | sme | nts | and | Proce | dures | ; | | | | | | | | |
| TB, HIV, HepB,<br>Hep C Ab, Anti-<br>CCP, Anti-<br>dsDNA, RF | Х | | | | | | | | | | | | | | | |
| FSH & estradiol (if applicable) | Х | | | | | | | | | | | | | | | |
| Serum<br>pregnancy test<br>(WCBP only) | X | | | | | | | | | | | | | | | |
| Urine pregnancy<br>test (WCBP<br>only) <sup>9</sup> | | X <sup>4</sup> | Х | Χ | | Χ | | X <sup>4</sup> | | Χ | | Х | | Χ | X | Χ |
| Haematology, chemistry, urinalysis | Х | X <sup>4</sup> | Х | Χ | | X <sup>10</sup> | | X <sup>4</sup> | | X <sup>10</sup> | | X <sup>10</sup> | | Χ | Х | Х |
| CRP | Χ | X <sup>4</sup> | | Χ | | Χ | | X <sup>4</sup> | | Χ | | Χ | | Χ | Χ | |
| Blood sample for PD inflammatory biomarkers, | | X <sup>4</sup> | | | | | | X <sup>4</sup> | | | | | | Χ | Х | |

| | 30) | | | | | | Trea | atment P | eriod <sup>1</sup> | 7 | | | | | wal <sup>18</sup> | -3)19 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening (-30) | Day 1 | Day 8 (±3) | Day 15 (±3) | Day 22 (±3) | Day 29 (±3) | Day 36 (±3) | <b>Day 43 (±3)</b><br>(week 6) | Day 50 (±3) | Day 57 (±3) | Day 64 (±3) | Day 71 (±3) | Day 78 (±3) | <b>Day 85 (+2)</b> (week 12) | Early Withdrawal <sup>18</sup> | Follow Up (±3)¹ <sup>9</sup> |
| mRNA, and TE <sup>11</sup> | | | | | | | | | | | | | | | | |
| PK blood<br>samples<br>GSK2982772 <sup>12</sup> | | Χ | X<br>4 | | | | | X <sup>4</sup> | | | | | | Х | X | |
| PK blood<br>samples for<br>MTX <sup>13</sup> | | X <sup>4</sup> | X<br>4 | | | | | X <sup>4</sup> | | | | | | | | |
| Pharmacogeneti c sample (PGx) | | X <sup>14</sup> | | | | | | | | | | | | | | |
| Synovial<br>biopsies for PK,<br>inflammatory<br>biomarkers,<br>mRNA, target<br>engagement &<br>pathway<br>engagement<br>analysis <sup>15</sup> | | X <sup>4,2</sup> 0 | | | | | | X4,21 | | | | | | | X <sup>16</sup> | |

#### Footnotes:

- 1. Full medical history (includes past and current conditions, medication history, substance usage, and family history of premature CV disease).
- 2. Full physical exam (includes height/weight at screening, height not measured at later time points).
- 3. Triplicate ECG to be performed at screening only.
- Pre-dose.
- 5. Any SAEs assessed as related to study participation (e.g., protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product will be recorded from the time a subject consents to participate in the study up to and including any follow-up. AEs will be collected from the start of Study Treatment until the follow-up contact. On Days 22, 36, 50, 64, and 78, subjects will be questioned about their general health status via phone call.
- All PRO assessments should be conducted on site before any tests, procedures, or assessments, to avoid influencing the subjects' perception.
- 7. DCE-MRI will be performed on all subjects, provided that sites have DCE-MRI capability and experience (e.g., hardware and software requirements). If sites do not have DCE-MRI capability or experience, a regular MRI will be performed of the affected hand/wrist. If the same joint is used for MRI and synovial biopsy, MRI should be performed before biopsy (if applicable).
- 8. Subjects must take study medication three times a day approximately 8 hours apart. Exact time of dosing to be recorded in diary cards. On Day 1, the first study dose will be administered at the site. On Days 8, 43 and 85 only, subjects must not take their medication at home in the morning. Subjects will complete pre-dose assessments and then will be administered their morning dose of medication at site on Days 8 and 43. On Day 85, subjects are no longer receiving study medication.
- 9. If urine pregnancy test is positive, a confirmatory serum pregnancy test must be performed.
- 10. Haematology and chemistry only. No urinalysis required on Days 29, 57 and 71. When clinical laboratory samples are taken on the same day as the MRI, the samples should be taken first prior to the administration of the contrast fluid with MRI. If this is not feasible (i.e. MRI is performed first), it is recommended that a separate IV catheter or straight venipuncture be performed in the *opposite* arm to where the MRI contrast fluid was administered.

- 11. Blood samples for inflammatory biomarkers, mRNA and target engagement. See laboratory manual for full details on sample collection, handling and shipment.
- 12. PK blood samples for GSK2982772 will be taken pre-dose on Days 8 and 43. Post-dose serial PK samples will be taken on Days 1, 8 and Day 43 at the following time points: 1, 2, 4, and 6 hours. A trough PK sample will be taken on Day 85 or at Early Withdrawal.
- 13. Only applicable if subjects are on MTX: PK blood samples for MTX will be taken pre-dose GSK2982772 on Day 1 (MTX alone), on Days 8 and 43 (MTX + GSK2982772). Subjects who are on MTX should ideally take their MTX dose on the same day of the week at approximately the same time of the day throughout the study. In addition, the Day 1, 8 and 43 visits should ideally be on the same day of the week.
- 14. A PGx blood sample is collected at the baseline visit, after the subject has been randomised and provided informed consent for genetic research. If the sample is not collected at the baseline visit, it can be collected at any time during the study after randomisation.
- 15. Synovial biopsies are optional.
- 16. Biopsy (if applicable) and MRI only are required at Early Withdrawal visit if subject withdraws after at least 14 days of treatment and prior to Day 43. If a subject withdraws between Days 43 and 57, an MRI is not required at the Early Withdrawal visit. If a subject withdraws on Day 57 or after, an MRI should be performed at the Early Withdrawal visit. A window allowance of ± 3 days of Early Withdrawal visit is allowed to perform the MRI.
- 17. Visit windows during the treatment period are relative to Day 1.
- 18. If a subject withdraws from the study, every effort will be made for the subject to complete an Early Withdrawal visit prior to the Follow Up visit.
- 19. Follow-up visit should be completed 28 days (±3 days) after the last dose of study medication.
- 20. MRI (and if applicable; a biopsy) may be performed during the screening window as an additional visit (if required) up to 7 days before Day 1 to allow sites flexibility in scheduling. The MRI must be completed prior to synovial biopsy (if performed on the same joint). The site should be reasonably confident that the subject has fully qualified for the study (e.g., screening clinical labs, vital signs, physical examination, etc.) before the MRI (and if applicable: a biopsy) is/are performed.
- 21. A biopsy (if applicable) and MRI may be performed on a separate day within the Day 43 window allowance (±3 days). A separate visit to perform the MRI followed by synovial biopsy (if applicable) is only allowed to accommodate scheduling. If biopsy is being performed, this visit must be scheduled after the Day 43 visit where the PK, clinical laboratory tests and other required Day 43 procedures are performed. Subjects must not take their study medication at home in the morning before the full Day 43 visit and also the morning before MRI and biopsy (if applicable) visit if being done on a separate day.
- 22. For MRI performed on day 85, a visit window of up to 2 days after is allowed in order to perform the MRI.

## 12.3. Appendix 3: Assessment Windows

## 12.3.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment unless otherwise specified. Treatment phases are to be included on A&R datasets.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date +1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

## 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |
| Post-Treatment | Any medication that is started >= Study Treatment Stop Date +1 |

#### 1. NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 12.4.2. Treatment Emergent Flag for Adverse Events

#### **Treatment States for AE Data**

| Treatment State | Definition |
|---|---|
| AE = Pre-Treatment | AE Start Date < Study Treatment Start Date |
| AE = On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date +1. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date +1 |
| AE = Post-Treatment | If AE onset date is after the treatment stop date+1. |
| | AE Start Date > Study Treatment Stop Date +1 |
| AE Onset Time | If Treatment Start Date > AE Onset Date: |
| Since 1st Dose | = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date ≤ AE Onset Date: |
| | = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| AE Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| AE = Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

• If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supply | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server UK1SALX00175 | |
| HARP Area | arenv \ arprod \ gsk2982772 \ mid203168 \ final |
| QC Spreadsheet | arenv \ arwork \ gsk2982772 \ mid203168 \ final \ documents |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Integrated Data Standards Library (IDSL) GSK<br/>A&amp;R dataset standards.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be | RTF files will be generated for all tables at the time of the SAC. |

## 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
• Subject level listings will not be provided in the main body of the GSK Clinical Study Report. All subject level listings will be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
- All unscheduled visits will be listed.

# Descriptive Summary Statistics Continuous Data Refer to IDSL Statistical Principle 6.06.1 Categorical Data N, n, frequency, %

#### **Graphical Displays**

• Refer to IDSL Statistical Principals 7.01 to 7.13.

Placebo in graphs to be shown in Blue and GSK2982772 in Red

```
style graphdata1/ color=BLUE contrastcolor=BLUE
linestyle=1 markersymbol="circlefilled";
    style graphdata2/ color=RED contrastcolor=RED
linestyle=34 markersymbol="trianglefilled";
```

For outputs which are displayed for all 4 treatment groups (ie by regimen)

## 12.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical | Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be | Not applicable |
| Derived by | |
| Programmer | |

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 12.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visit (including
  unscheduled visits) for safety parameters will be counted in both the High and Low categories of "Any
  visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential
  Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 12.6.2. Study Population

## **Demographics**

#### Date of Birth

Only the year of birth will be captured, and therefore the date of birth is then derived as follows:
 Year of birth = YYYY → Date of birth = PPD YYYY

#### Age

- Calculated as the integer part of (date of screening date of birth)
   Age = integer part (date of screening PPD YYYYY)
- Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### Race category

- White: 'White: Arabic/North African Heritage' and 'White: White/Caucasian/European Heritage', or both of these, but no other category checked
- African descent: 'African American/African Heritage', and no other category checked
- Asian: 'Asian Central/South Asian Heritage', 'Asian East Asian Heritage', 'Asian Japanese Heritage', and 'Asian – South East Asian Heritage', or any combination of these, but no other category checked
- Other: Any combination that has not been categorized above ('mixed race')

#### Disease **History**

Time since formal diagnosis= date of visit - date of formal diagnosis-

Time since onset of first musculoskeletal symptoms= date of visit - date of first musculoskeletal symptoms-

## **Demographics**

If date of visit is missing use screening date.

#### **Treatment Compliance**

- Subject compliance will be based on the number of expected tablets to be taken and the number actually taken and will depend on whether a subject was taking investigational product (two 30mg tablets) twice a day or three times according to the regimen they were randomized to:
  - Total tablets taken is (Total number of Tablets Dispensed-Total Tablets Returned)
  - Duration of exposure is calculated as described in extent of exposure section below
  - Total Tablets expected to be taken is duration of exposure\*4 for BID subjects and \*6 for TID subjects

Note: if any of the tablets dispensed/returned contain missing number of tablets total tablets taken will be set to missing.

• Treatment compliance will be calculated based on the formula:

Treatment Compliance = (Total tablets taken/total tablets expected to be taken)\*100

#### where

Note compliance will only be calculated for subjects who took at least one dose (i.e.) number of tablets taken is >=1

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

Cumulative Dose = Total Tablets taken\*30 for GSK2982772 subjects

Cumulative dose will be 0 for placebo subjects.

Note: If the total tablets taken is missing cumulative dose will be set to missing.

## 12.6.3. **Efficacy**

## 12.6.3.1. HAQ-DI

The functional status of the subject will be assessed by means of the Disability Index of the Stanford Health Assessment Questionnaire (HAQ-DI). This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas:

• dressing & grooming, rising, eating, walking, hygiene, reach, grip, and common daily activities.

Each functional area contains at least two questions. For each question, there is a four-level response set that is scored from 0 (without any difficulty) to 3 (unable to do). If aids or devices or physical assistance are used for a specific functional area and the maximum response of this functional area is 0 or 1 the according value is increased to a score of 2.

#### **HAQ-DI Aids**

| Aid or equipment | Will be associated with category score |
|---|---|
| Walking stick/frame, crutches, wheelchair | Walking |
| Aids used for dressing | Dressing and grooming |
| Specially adapted utensils | Eating |
| Specially adapted chair | Rising |
| Raised toilet seat, bath rail, bath seat | Hygiene |
| Long-handled appliance in bathroom | Hygiene |
| Long-handled appliance for reaching | Reach |
| Jar opener | Grip |
| Other (1) | Dressing & grooming, rising, eating, walking |
| Other (2) | hygiene, reach, grip, common daily activities |

If "other" is marked as an aid or equipment, then this can be assigned to a group of four functional areas and will be handled as an aid or equipment for each of the four functional areas. Therefore, if the maximum score of a functional area is 0 or 1 that value is increased to a score of 2 for each of the four functional areas.

Regarding these corrections, the highest response within each functional area determines the score of that specific functional area. If no questions within a given functional area were answered, no score will be provided for that category (even if answers on aids or equipment are available).

HAQ-DI is only calculated if there are at least 6 functional area scores available.

The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. If there are less than 6 functional area scores available, no imputation will be done and the HAQ-DI will be set to missing for the according assessment.

#### 12.6.3.2. Patient Global Assessment

The patient global assessment of arthritis disease activity (PtGA) is measured on a 10cm visual analogue scale (VAS) with values 0=very well to 10=very poor. More commonly this measurement is reported as measured off the 10cm VAS in mm. For reporting purposes, the VAS measurement from the eCRF will be converted from cm to mm by multiplying values by 10. All listings and summaries of the PtGA will be using mm.

## 12.6.3.3. Physician Global Assessment (PGA)

The physician global assessment of arthritis disease activity (PGA) is measured on a 10cm visual analogue scale (VAS) with values 0=none to 10=extremely active. More commonly this measurement is reported as measured off the 10cm VAS in mm. For reporting purposes, the VAS measurement from the eCRF will be converted from cm to mm by multiplying values by 10. All listings and summaries of the PGA will be using mm.

#### 12.6.3.4. Disease Activity Score (DAS28):

Disease activity Score (DAS28 CRP) is a numeric outcome based on Tender joint count 28 (TJC28), swollen joint count 28 (SJC28), C-reactive protein (CRP) and patient global assessment (PtGA). CRP values will be taken from the clinical chemistry data within the lab dataset.

The joint counts will be based on 28 joints as follows (both left and right sides): Shoulder, elbow, wrist, metacarpophalangeal (first (thumb), second, third, fourth, fifth), proximal interphalangeal (thumb (interphalangeal), index, middle, ring, little) and knee.

The DAS28-CRP score will be calculated using the following formula:

DAS28 - CRP = 
$$0.56 * \sqrt{TJC28} + 0.28 * \sqrt{SJC28} + 0.36 * \ln(CRP + 1) + 0.014$$
  
\* PtGA + 0.96.

- If one of the components is missing at an individual assessment point, the DAS28-CRP value for that assessment will be set to missing.
- Note PtGA must be measured in mm for this calculation as described in Section 12.6.3.2

## Categorical DAS28 Response

DAS28-CRP scores will each be categorized using EULAR response criteria. Response at a given time point is defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to baseline. The definition of no response, moderate response and good response is captured in the following table:

| Table 4 | <b>EULAR Response Criteria</b> |
|---------|--------------------------------|
|---------|--------------------------------|

| Current | DAS28 decrease from baseline value | | | DAS28 decrease from baseline value |
|---|---|---|---|---|
| DAS28 | >1.2 $>0.6 \text{ to } \le 1.2$ $\le 0.6$ | | | |
| ≤ 3.2 | Good response | Moderate response | No response | |
| $> 3.2 \text{ to} \le 5.1$ | Moderate response | Moderate response | No response | |
| > 5.1 | Moderate response | No response | No response | |

If the post-baseline DAS28-CRP score is missing, then the corresponding EULAR category will be missing. If the baseline DAS28-CRP is missing, then all post-baseline EULAR response values will be missing.

## DAS28 Low Disease Activity (LDA)

DAS28-CRP Low Disease Activity is defined as a DAS28 score of <3.2.

#### DAS28 Remission

DAS28-CRP remission is achieved by a DAS28-CRP value <= 2.6.

## 12.6.3.5. ACR Response Rates

The American College of Rheumatology's (ACR) definition for calculating improvement in RA is calculated as a 20% improvement (ACR20) in both tender and swollen joint counts and 20% improvement in at least 3 of the 5 remaining ACR-core set measures: patient and physician global assessments, patient's assessment of arthritis pain, disability (HAQ-DI), and an acute-phase reactant (i.e. CRP value). Similarly, ACR50 and ACR70 are calculated with the respective percent improvement. This efficacy measurement will be made at every post-baseline study assessment time point.

The specific components of the ACR Assessments that will be used in this study are as follows and can be grouped into three components:

- Tender/Painful Joint count (28)
- Swollen Joint Count (28)
- 5 Remaining ACR-Core Set Measures:
  - Patient Assessment of Joint Pain
  - PtGA

- PGA
- CRP
- HAQ-DI

For all visits, if any of the component scores are missing, meaning ACR20/50/70 responder definitions cannot be properly assessed, then those scores will be considered as not having met the criteria for improvement. Therefore, if TJC28 or SJC28 or 3 or more of the 5 remaining ACR-core set measures are missing, ACR20/ ACR50/ ACR70 will each be considered as "no response" in the DAS\_ACR dataset.

For missing Baseline values or a Baseline value of 0, the percentage improvement can't be calculated and the ACR will be considered as not having met the criteria for improvement

e.g.

- if TJC28 or SJC28 is missing or 0 at baseline then ACR20/50/70 will be considered as 'no response'
- if TJC28 and SJC28 are non-missing and >0 at baseline but there are < 3 of the 5 remaining core set measures that are non-missing and >0 at baseline then ACR20/50/70 will be considered as 'no response'

Data from the screening visit will not be used to impute baseline.

## 12.6.3.6. Swollen and Tender/Painful Joint Count

Four different scores will be calculated to evaluate swelling and tenderness of joints. TJC28 and SJC28 will take 28 joints into account.

The assessment for swelling is the total number of joints with a present swelling and ranges from 0 to 28 for SJC28.

The assessment for tenderness is the total number of joints with a present tenderness and ranges from 0 to 28 for TJC28.

The following 28 joints will be taken into account for TJC28 and SJC28: Shoulder (2 joints), Knee (2), Elbow (2), Wrist (2), Fingers (PIP, MCP: 20).

Artificial, ankylosed and missing joints are excluded from swelling and tenderness assessment.

If there are missing or excluded observations for tender or swollen joints then the remaining observations will be assessed and weighted by dividing the number presented by number of non-missing and by multiplying by 28 for the joint count. No imputations for individual joints will be done. If a joint is not evaluable at Baseline, then that joint is set to missing throughout the study.

If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.

Observed joint states will be listed without any modification for every subject and visit.

#### 12.6.3.7. FACIT-Fatigue

The FACT-G scoring guide identifies those items which must be reversed before being added to obtain subscale totals. Items are scored using a Likert scale from 0 to 4, to "0" (not at all) to "4" (very much).

In order to calculate a total score negatively stated items are reversed by subtracting the response from "4". After reversing proper items, all subscale items are summed to a total, which is the subscale score. For all FACIT scales and symptom indices, the higher the score the better the QOL.

Negatively stated items refer to all statements asked except ('I have energy' and 'I am able to do my usual activities')

Fatigue Score =  $[\text{sum of Item Scores}] \times [13] / [\text{number of items answered}].$ 

A Fatigue score will only be calculated if at least 7 responses have been provided.

#### 12.6.3.8. DCE-MRI

Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) parameters are measured at each individual joint and consist of:

- Exchange Rate (K<sup>trans</sup>)
- Interstitial Volume (V<sub>e</sub>)
- Plasma Volume (V<sub>p</sub>)
- Initial Rate of Enhancement (IRE)
- Maximum signal intensity enhancement (ME).

All DCE-MRI parameters will be presented as a total measure over all joints at each time point.

DCI-MRI parameters will be calculated as:

$$\frac{\sum_{all\ joints}(Parameter)}{Number\ of\ Joints}$$

Parameters will also be presented normalized by the VEP.

Normalized DCE-MRI parameters will be calculated as:

$$\frac{\sum_{\textit{all joints}}(\textit{VEP} * \textit{Parameter})}{\sum_{\textit{all joints}}\textit{VEP}}$$

If parameters are missing for individual joints, these joints will be excluded from the numerator and denominator of the calculation.

If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit. This threshold might be altered after review of the actual raw data.

## 12.6.3.9. CDAI and SDAI

Although not specified in the protocol as endpoints both the Simple Disease Activity Index (SDAI) and clinical disease activity index (CDAI) will be calculated and summarised.

#### SDAI

SDAI is a composite score calculated using the formula:

Where PtGA and PGA is measured 0-10 and CRP is measured in (mg/dl). Higher values represent higher disease activity.

If one of the components is missing at an individual assessment point, the SDAI value for that assessment will be set to missing.

**SDAI** Remission

SDAI <= 3.3

SDAI Low Disease Activity 3.3 < SDAI <= 11

## **CDAI**

CDAI is a composite score calculated using the following formula:

CDAI= SJC28+ TJC28 + PtGA+ PGA

Where PtGA and PGA are measured 0-10. CDAI ranges from 0 to 76 with higher values representing higher disease activity.

Remission is achieved for a non-missing CDAI value ≤2.8 and

Low Disease Activity 2.8 < CDAI <= 10

If one of the components is missing at an individual assessment point, no imputations will be done and the CDAI value for that assessment will be set to missing.

## 12.6.4. Safety

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1

#### **ECG Parameters**

#### RR Interval

IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### 12.6.5. Biomarker

#### **TEAR**

## **Target Engagement**

- Ratio = free / total
- Target Engagement = 100 (ratio post/ratio baseline) \* 100))
- BIOMARK dataset:

BICAT = TRIPK1 (total) or FRIPK1 (free) for the same smpty

#### 12.6.6. PK

Synovial Tissue Pharmacokinetic Concentrations

#### Synovial Tissue PK Conc

- The density of human synovial tissue is 1.184 g/mL per Gastroplus V9.0.
- The volume of solvent added to each tissue sample was 0.5 mL.
- For actual tissue weights, please refer to the Excel spreadsheet

#### Synovial PK Concentration (ng/mL)

- 1. PK Conc in Weight of Tissue Sample = SMS PK Conc in Soln (ng/mL) X [0.5 mL + (Tissue Weight (g) / 1.184 g/mL)]
- 2. PK Conc in tissue as concentration (ng/g) = PK Conc in Weight of Tissue Sample / Tissue Weight
- 3. PK Conc in tissue as concentration (ng/mL) = PK Conc in tissue as concentration (ng/g) 1.184 g/mL

Example (fictitious) data:

SMS tissue homogenate concentration = 2 ng/mL

Tissue weight = 0.014 g

SMS plasma concentration= 400 ng/mL

**Example Calculations:** 

- 1. Convert GSK2982772 concentration in the homogenate to GSK2982772 concentration in the tissue sample as follows:
- 2 ng/mL X  $[0.5 \text{ mL} + (0.014 \text{ g/1.184 g/mL})] = 2 \text{ng/mL} \times 0.512 \text{ mL} = 1.024 \text{ ng GSK2982772 in a} 0.014 g tissue sample$
- 2. Convert absolute amount of GSK2982772 in this skin tissue sample to a tissue concentration as follows:
- 1.024 ng / 0.014 g tissue = 73.1 ng GSK2982772/g tissue = 73.1 ng/g
- Convert ng/g tissue to ng/mL tissue as follows:
- 73.1 ng/g X 1.184 g/mL = 86.5 ng GSK2982772/mL tissue = 86.5 ng/mL
- 4. Determine the ratio of GSK2982772 tissue concentration to GSK2982772 plasma concentration for a given patient as follows:
- 86.5 ng/mL / 400 ng/mL = 0.216

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion was defined as one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study at the discretion of the investigator.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. Withdrawal visits will not be summarised and will be listed only.</li> </ul> |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be |
| | documented along with the reason for exclusion in the clinical study report. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> </ul> |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

# 12.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Deticat | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | l | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 12.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | · · | | |
| | | > 450 | < 480 |
| Absolute QTc Interval | msec | ≥ 480 | <500 |
| | | ≥ 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 30 | ≤ 59 |
| increase from Daseline Q10 | msec | ≥ 60 | |

# 12.8.3. Vital Signs

| Vital Sign Parameter Units | | Clinical Concern Range | |
|----------------------------|------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | Bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease In | | Incre | crease |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | Bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

# 12.9. Appendix 11: Abbreviations & Trade Marks

# 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACR | American College of Rheumatology |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CARLOS | Cartilage Loss Scoring System |
| CDAI | Clinical Disease Activity Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRP | C-reactive protein |
| CS | Compound symmetry |
| CSH | Heterogenous compound symmetry |
| CSR | Clinical Study Report |
| CV | Cardiovascular |
| CV <sub>b</sub> | Coefficient of Variation (Between) |
| DAS 28-CRP | Disease Activity Score 28-CRP |
| DBF | Database Freeze |
| DBR | Database Release |
| DCE-MRI | Dynamic Contrast-Enhanced Magnetic Resonance Imaging |
| DOB | Date of Birth |
| DP | Decimal Places |
| DRC | Data Review Committee |
| DVT | Deep vein thrombosis |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GCSP | Global Clinical Safety & Pharmacovigilence |
| GSK | GlaxoSmithKline |
| HAQ-DI | Disability Index of the Stanford Health Assessment Questionnaire |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| II | Immuno-Inflammation |
| IRE | Initial rate of enhancement |
| Ktrans | Exchange rate |
| LS | Least squared |
| ME | Maximal signal intensity enhancement |
| MMRM | Mixed Model Repeated Measures |
| MRI | Magnetic Resonance Imaging |
| MTX | Methotrexate |

| Abbreviation | Description |
|---|---|
| OMERACT- | Outcome Measures in Rheumatology, Rheumatoid Arthritis Magnetic |
| RAMRIS | Resonance Image Scoring System |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PE | Pulmonary embolism |
| PGA | Physician Global Assessment |
| PK | Pharmacokinetic |
| PK772 | Pharmacokinetic GSK298772 |
| PKMeth | Pharmacokinetic Methotrexate |
| PP | Per Protocol |
| PopPK | Population PK |
| PtGA | Patient Global Assessment |
| QC | Quality Control |
| QOL | Quality of Life |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RA | Rheumatoid Arthritis |
| RAMOS | Randomization & Medication Ordering System |
| RAMRIQ | Rheumatoid Arthritis MRI Quantitative |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SDAI | Simple Disease Activity Index |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SJC28 | Swollen Joint Count 28 |
| SRT | Safety Review Team |
| TA | Therapeutic Area |
| TEAR1 | Target Engagement Assay RIP1 |
| TIA | Transient ischemic attack |
| TFL | Tables, Figures & Listings |
| TJC28 | Tender Joint Count 28 |
| VAS | Visual Analogue Scale |
| Ve | Interstitial volume |
| Vep | Volume of enhancing Pannus |
| $V_p$ | Plasma volume |

# 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

ADVAIR

| Trademarks not owned by the |
|-------------------------------------------|
| <b>GlaxoSmithKline Group of Companies</b> |

NONMEM

SAS

WinNonlin

## 12.10. Appendix 12: List of Data Displays

## 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|-----------------|-------------|
| Study Population | 1.1 to 1.18 | NA |
| Efficacy | 2.1 to 2.67 | 2.1 to 2.23 |
| Safety | 3.1 to 3.24 | 3.1 to 3.3 |
| Pharmacokinetic | 4.1 to 4.2 | 4.1 to 4.7 |
| Pharmacokinetic / Pharmacodynamic | NA | 5.1 to 5.3 |
| Biomarker | 6.1 to 6.14 | 6.1 to 6.7 |
| Section | Listi | ings |
| ICH Listings | 1 to 40, and 85 | |
| Other Listings | 41 to | o 84 |

# 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

## 12.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| AR | Administrative review, delivered by the GSK stats and programming team |
| SAC [1] | Final Statistical Analysis Complete responsibility of Quanticate |
| SAC2 [1] | Post SAC and delivered by the GSK stats and programming team |

#### NOTES:

<sup>•</sup> Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.10.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition for the Study Conclusion Record | ICH E3, FDAAA, EudraCT Add footnote: Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK Display Standards and CDISC SDTM/ADaM standards. | AR<br>SAC[1] |
| 1.2. | Safety | SD1 /<br>SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | AR<br>SAC[1] |
| 1.3. | All subjects | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC[1] |
| 1.4. | Randomised | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations Please add footnote to say that randomised population=enrolled population | SAC[1] |
| Protoco | Protocol Deviation | | | | |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC[1] |

| Study | Population Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | opulation Analysed | | | | |
| 1.6. | All subjects | SP1 | Summary of Study Populations | IDSL | SAC[1] |
| Demog | graphic and Bas | eline Characteris | tics | | |
| 1.7. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT Include summary of time since formal diagnosis of RA and time since onset of first musculoskeletal symptoms | SAC[1] |
| 1.8. | Randomised | DM11 | Summary of Age Ranges | EudraCT Please add footnote to say that randomised population=enrolled population | SAC[1] |
| 1.9. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC[1] |
| 1.10. | Safety | SU1 | Summary of Tobacco Use | IDSL | SAC[1] |
| Prior a | nd Concomitan | t Medications | | | |
| 1.11. | Safety | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC[1] |
| 1.12. | Safety | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC[1] |
| 1.13. | Safety | MH1 | Summary of Past Cardiovascular Risk Factors | ICH E3 Include only pre-defined list | SAC[1] |
| 1.14. | Safety | MH1 | Summary of Current Cardiovascular Risk Factors | ICH E3 Include only pre-defined list | SAC[1] |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.15. | Safety | FH1 | Summary of Family History: Cardiovascular Risk Factors | IDSL | SAC[1] |
| 1.16. | Safety | CM1 | Summary of Prior Medications | ICH E3 | AR<br>SAC[1] |
| 1.17. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 | AR<br>SAC[1] |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.18. | Safety | EX1 /<br>EX5 | Summary of Exposure to Study Treatment | ICH E3 | SAC[1] |

# 12.10.5. Efficacy Tables

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficac | У | | | | |
| 2.1. | Safety | EFF_T1 | Summary of FACIT-Fatigue by Visit | | AR<br>SAC [1] |
| 2.2. | Safety | EFF_T2 | Summary of Change from Baseline in FACIT-Fatigue by Visit | | AR<br>SAC [1] |
| 2.3. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in FACIT-Fatigue | | AR<br>SAC [1] |
| 2.4. | Safety | EFF_T1 | Summary of HAQ-DI by Visit | | AR<br>SAC [1] |
| 2.5. | Safety | EFF_T2 | Summary of Change from Baseline in HAQ-DI by Visit | | AR<br>SAC [1] |
| 2.6. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in HAQ-DI | | AR<br>SAC [1] |
| 2.7. | Safety | EFF_T1 | Summary of Patient Global Assessment by Visit | | SAC [1] |
| 2.8. | Safety | EFF_T2 | Summary of Change from Baseline in Patient Global Assessment by Visit | | SAC [1] |
| 2.9. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Patient Global Assessment | | SAC [1] |
| 2.10. | Safety | EFF_T1 | Summary of Physician Global Assessment by Visit | | SAC [1] |
| 2.11. | Safety | EFF_T2 | Summary of Change from Baseline in Physician Global Assessment by Visit | | SAC [1] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Physician Global Assessment | | SAC [1] |
| 2.13. | Safety | EFF_T1 | Summary of DAS28(CRP) by Visit | | AR<br>SAC [1] |
| 2.14. | Safety | EFF_T2 | Summary of Change from Baseline in DAS28(CRP) by Visit | | AR<br>SAC [1] |
| 2.15. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in DAS28(CRP) | | AR<br>SAC [1] |
| 2.16. | Safety | EFF_T1 | Summary of DAS28(CRP) by Visit and Dosing Regimen | Separate page for BID and TID | AR<br>SAC [1] |
| 2.17. | Safety | EFF_T2 | Summary of Change from Baseline in DAS28(CRP) by Visit and Dosing Regimen | Separate page for BID and TID | AR<br>SAC [1] |
| 2.18. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in DAS28(CRP) and Dosing Regimen | Separate page for BID and TID | AR<br>SAC [1] |
| 2.19. | Safety | EFF_T4 | DAS28-CRP EULAR Response Categories | | AR<br>SAC [1] |
| 2.20. | Safety | EFF_T4 | DAS28-CRP Remission and Low Disease Activity | Update column for EULAR response to be summarise number and percent of subjects meeting remission and LDA criteria by visit | AR<br>SAC [1] |
| 2.21. | Safety | EFF_T5 | ACR Response Rates by Visit | | AR<br>SAC [1] |
| 2.22. | Safety | EFF_T4 | DAS28-CRP EULAR Response Categories and Dosing Regimen | Separate page for BID and TID | AR<br>SAC [1] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | Safety | EFF_T4 | DAS28-CRP Remission and Low Disease Activity and Dosing Regimen | Separate page for BID and TID Update column for EULAR response to be summarise number and percent of subjects meeting remission and LDA criteria by visit | AR<br>SAC [1] |
| 2.24. | Safety | EFF_T5 | ACR Response Rates by Visit and Dosing Regimen | Separate page for BID and TID | AR<br>SAC [1] |
| 2.25. | Safety | EFF_T1 | Summary of Tender Joint Count (28 Joints) by Visit | | AR<br>SAC [1] |
| 2.26. | Safety | EFF_T2 | Summary of Change from Baseline in Tender Joint Count (28 Joints) by Visit | | AR<br>SAC [1] |
| 2.27. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Tender Joint Count (28 Joints) | | AR<br>SAC [1] |
| 2.28. | Safety | EFF_T1 | Summary of Swollen Joint Count (28 Joints) by Visit | | AR<br>SAC [1] |
| 2.29. | Safety | EFF_T2 | Summary of Change from Baseline in Swollen Joint Count (28 Joints) by Visit | | AR<br>SAC [1] |
| 2.30. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Swollen Joint Count (28 Joints) | | AR<br>SAC [1] |
| 2.31. | Safety | EFF_T1 | Summary of MRI parameters: RAMRIS scoring system | Separate page for each parameter | SAC [1] |
| 2.32. | Safety | EFF_T2 | Summary of Change from Baseline in MRI parameters: RAMRIS scoring system | Separate page for each parameter | SAC [1] |
| 2.33. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in MRI parameters: RAMRIS scoring system | Separate page for each parameter | SAC [1] |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | Safety | EFF_T1 | Summary of MRI parameters: RAMRIQ scoring system | Separate page for each parameter | SAC [1] |
| 2.35. | Safety | EFF_T2 | Summary of Change from Baseline in MRI parameters: RAMRIQ scoring system | Separate page for each parameter | SAC [1] |
| 2.36. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in MRI parameters: RAMRIQ scoring system | Separate page for each parameter | SAC [1] |
| 2.37. | Safety | EFF_T1 | Summary of MRI parameters: CARLOS scoring system | Separate page for each parameter | SAC [1] |
| 2.38. | Safety | EFF_T2 | Summary of Change from Baseline in MRI parameters: CARLOS scoring system | Separate page for each parameter | SAC [1] |
| 2.39. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in MRI parameters: CARLOS scoring system | Separate page for each parameter | SAC [1] |
| 2.40. | Safety | EFF_T1 | Summary of synovial inflammation DCE-MRI | Separate page for each parameter | SAC [1] |
| 2.41. | Safety | EFF_T2 | Summary of Change from Baseline in synovial inflammation DCE-MRI | Separate page for each parameter | SAC [1] |
| 2.42. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in synovial inflammation DCE-MRI | Separate page for each parameter | SAC [1] |
| 2.43. | Safety | EFF_T1 | Summary of synovial inflammation DCE-MRI by Dosing Regimen | Separate page for each parameter/Dosing regimen | SAC [1] |
| 2.44. | Safety | EFF_T2 | Summary of Change from Baseline in synovial inflammation DCE-MRI by Dosing Regimen | Separate page for each parameter/Dosing regimen | SAC [1] |
| 2.45. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in synovial inflammation DCE-MRI by Dosing Regimen | Separate page for each parameter/Dosing regimen | SAC [1] |
| 2.46. | Safety | EFF_T1 | Summary of Patient Assessment of joint Pain by Visit | | AR<br>SAC [1] |
| 2.47. | Safety | EFF_T2 | Summary of Change from Baseline in Patient Assessment of joint pain by Visit | | AR<br>SAC [1] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.48. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Patient Assessment of joint pain | | AR<br>SAC [1] |
| 2.49. | Safety | DM1 | Summary of RA symptom Questionnaire | Add column for visit Summary statistics for numeric responses and number (%) in each category for each other question | SAC [1] |
| 2.50. | Safety | EFF_T1 | Summary of CRP by Visit | | SAC [1] |
| 2.51. | Safety | EFF_T2 | Summary of Change from Baseline in CRP by Visit | | SAC [1] |
| 2.52. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in CRP | | SAC [1] |
| 2.53. | PP | EFF_T1 | Summary of DAS28(CRP) by Visit | | SAC [1] |
| 2.54. | PP | EFF_T2 | Summary of Change from Baseline in DAS28(CRP) by Visit | | SAC [1] |
| 2.55. | PP | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in DAS28(CRP) | | SAC [1] |
| 2.56. | PP-<br>completer | EFF_T1 | Summary of DAS28(CRP) by Visit-Per protocol Completers | Include subjects who completed the study and are in PP population | SAC [1] |
| 2.57. | PP-<br>completer | EFF_T2 | Summary of Change from Baseline in DAS28(CRP) by VisitPer protocol Completers | Include subjects who completed the study and are in PP population | SAC [1] |
| 2.58. | PP-<br>completer | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in DAS28(CRP)Per protocol Completers | Include subjects who completed the study and are in PP population | SAC [1] |
| 2.59. | Safety | EFF_T1 | Summary of Clinical Disease Activity Index by Visit | | AR<br>SAC [1] |
| 2.60. | Safety | EFF_T2 | Summary of Change from Baseline in Clinical Disease Activity Index by Visit | | AR<br>SAC [1] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.61. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Clinical Disease Activity Index | | AR<br>SAC [1] |
| 2.62. | Safety | EFF_T1 | Summary of Simple Disease Activity Index by Visit | | AR<br>SAC [1] |
| 2.63. | Safety | EFF_T2 | Summary of Change from Baseline in Simple Disease Activity Index by Visit | | AR<br>SAC [1] |
| 2.64. | Safety | EFF_T3 | Summary of Statistical Analysis Results for Change from Baseline in Simple Disease Activity Index | | AR<br>SAC [1] |
| 2.65. | Safety | EFF_T6 | Summary of Bayesian Analysis of Change from Baseline in DAS28-CRP at day 85 | GSK Responsibility<br>seed=5235 thin=50<br>nbi=1000 nmc=500000 | AR<br>SAC [1] |
| 2.66. | Safety | EFF_T7 | Summary of Bayesian Analysis of ACR20 at day 85 | GSK Responsibility Seed=240, nbi=1000 nmc=100000 thin=10 | AR<br>SAC [1] |
| 2.67. | Safety | EFF_T7 | Summary of Bayesian Analysis of ACR50 at day 85 | GSK Responsibility Seed=241, nbi=1000 nmc=100000 thin=10 | AR<br>SAC [1] |

Note for MRI parameters, a list of expected bones/joints for DCE and RAMRIS can be provided in an excel file on request.

# 12.10.6. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficac | y | | | | |
| 2.1. | Safety | EFF_F1 | FACIT-Fatigue, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.2. | Safety | EFF_F1 | HAQ-DI, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.3. | Safety | EFF_F1 | Patient Global Assessment, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | SAC [1] |
| 2.4. | Safety | EFF_F1 | Physician Global Assessment, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | SAC [1] |
| 2.5. | Safety | EFF_F1 | DAS28-CRP, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.6. | Safety | EFF_F2 | Individual Subject Profiles for DAS28-CRP | | SAC [1] |
| 2.7. | Safety | EFF_F1 | DAS28-CRP, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment and Dosing regimen over Time | Separate page for each dosing regimen | AR<br>SAC [1] |
| 2.8. | Safety | EFF_F3 | Proportion (± SE) of subjects in each DAS28-CRP EULAR Response Category | Separate page for each EULAR response category | AR<br>SAC [1] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | Safety | EFF_F4 | Proportion (±SE) of subjects achieving ACR20/50/70 | Separate page for AC20/50 and 70 | AR<br>SAC [1] |
| 2.10. | Safety | EFF_F1 | Tender Joint Count (28), Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.11. | Safety | EFF_F1 | Swollen Joint Count (28), Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.12. | Safety | EFF_F1 | MRI parameters: RAMRIS scoring, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Separate page for each parameter | SAC [1] |
| 2.13. | Safety | EFF_F1 | MRI parameters: RAMRIQ scoring, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Separate page for each parameter | SAC [1] |
| 2.14. | Safety | EFF_F1 | MRI parameters: CARLOS scoring, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Separate page for each parameter | SAC [1] |
| 2.15. | Safety | EFF_F1 | DCE-MRI, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Separate page for each parameter | SAC [1] |
| 2.16. | Safety | EFF_F2 | Individual Subject Profiles for DCE-MRI | Separate page for each parameter | SAC [1] |
| 2.17. | Safety | EFF_F1 | DCE-MRI, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment and Dosing Regimen over Time | Separate page for each parameter/dosing regimen | SAC [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | Safety | EFF_F1 | Patient Assessment of Joint Pain, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Separate page for each parameter | AR<br>SAC [1] |
| 2.19. | Safety | EFF_F1 | CRP, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.20. | PP | EFF_F1 | DAS28-CRP, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | SAC [1] |
| 2.21. | PP-<br>Completer | EFF_F1 | DAS28-CRP, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | Include subjects who completed the study and are in PP population | SAC [1] |
| 2.22. | Safety | EFF_F1 | Clinical Disease Activity Index, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |
| 2.23. | Safety | EFF_F1 | Simple Disease Activity Index, Adjusted Mean (±SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | AR<br>SAC [1] |

# 12.10.7. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | [Safety] | AE1 | Summary of Adverse Events by System Organ Class and Preferred Term | IDSL | SAC [1] |
| 3.2. | [Safety] | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term | ICH E3 | SAC [1] |
| 3.3. | [Safety] | AE3 | Summary of Common (≥10%) Adverse Events by Overall Frequency | ICH E3 Common defined as >= 10% within either treatment group | SAC [1] |
| 3.4. | [Safety] | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 | SAC [1] |
| 3.5. | [Safety] | AE15 | Summary of Common (≥10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | SAC [1] |
| 3.6. | [Safety] | AE3 | Summary of Common (≥10%) Drug-Related Adverse Events by Overall Frequency | ICH E3 | SAC [1] |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 3.7. | [Safety] | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | SAC [1] |
| 3.8. | [Safety] | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency | IDSL | SAC [1] |

| Safety: Tables | | | | |
|---|---|---|---|---|
| No. Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events | FDAAA, EudraCT | SAC [1] |
| Laboratory: Chemistr | у | | | |
| 3.10. [Safety] | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC [1] |
| 3.11. [Safety] | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | SAC [1] |
| 3.12. [Safety] | LB17 | Summary of Worst Case Lipids Results by NR Criteria Post-Baseline Relative to Baseline by Randomised Treatment | ICH E3 (i.e. treatment emergent) Lipids parameters = LDL, HDL Recommended for larger studies, could be covered by listings for smaller studies. The specific criteria to be defined by the study/project team. Values could be categorized by: [1] Above/below reference range (e.g., normal range, clinical concern range). [2] Graded toxicity scales. [3] Changes from baseline to reference range category. Or [1] On-treatment. [2] Post-baseline (i.e., anything after first dose and not necessarily while Ontreatment). [3] Through IP end + X days, etc. | SAC [1] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | [Safety] | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC[1] |
| 3.14. | [Safety] | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | SAC[1] |
| Labora | tory: Urinalysis | ; | | | |
| 3.15. | [Safety] | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 | SAC[1] |
| 3.16. | [Safety] | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | SAC[1] |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.17. | [Safety] | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC[1] |
| 3.18. | [Safety] | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC[1] |
| ECG | | | | | |
| 3.19. | [Safety] | EG1 | Summary of ECG Findings | IDSL | SAC[1] |
| 3.20. | [Safety] | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC[1] |
| 3.21. | [Safety] | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC[1] |
| 3.22. | [Safety] | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC[1] |
| Vital Si | gns | | | | |
| 3.23. | [Safety] | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC[1] |
| 3.24. | [Safety] | VS7 | Summary of Worst Case Vital Signs by PCI Criteria Post-<br>Baseline Relative to Baseline | IDSL | SAC[1] |

# 12.10.8. Safety Figures

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events | | | | |
| 3.1. | [Safety] | AE10 | Plot of Common (≥10%) Adverse Events and Relative Risk | IDSL | SAC[1] |
| Laborat | ory | | | | |
| 3.2. | [Safety] | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | IDSL | SAC[1] |
| 3.3. | [Safety] | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | IDSL | SAC[1] |

# 12.10.9. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | PK Concentration | | | | |
| 4.1. | PK772 | PK01 | Summary of Plasma GSK2982772 Concentration-Time Data (ng/mL) by Dosing Regimen | Pre-dose, Day 1, 8, 43 and 85. Day 1, 8 and 43 at 1, 2, 4 and 6 h post dose | AR<br>SAC [1] |
| 4.2. | PKMeth | PK01 | Summary of Plasma Methotrexate Concentration Data (ng/mL) by Dosing Regimen | Pre-dose Day 1, 8 and 43 | SAC[1] |

# 12.10.10. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Concentration | | | | | |
| 4.1. | PK772 | PK_F1 | Spaghetti plot of GSK2982772 Individual Plasma Concentration Data by Study Day | Spaghetti plot of individual trough concentrations vs day (8, 43 and 85). Separate panels for each per regimen (bid and tid) | SAC [1] |
| 4.2. | PK772 | PK_F2 | GSK2982772 Trough Plasma Concentration Data by Study Day | Plot of individual trough concentrations vs day (8, 43 and 85) and overlaid with box and whisker plot. Separate panels for each regimen (bid and tid) | AR<br>SAC [1] |
| 4.3. | PK772 | PK_F3 | GSK2982772 Plasma Concentration Data by time relative to dose | Spaghetti plot of observed plasma concentration versus time (pre-dose =0, 1, 2, 4, and 6 hours post dose). One panel for each regimen and separate pages for each day (1, 8, and 43) | AR<br>SAC [1] |
| 4.4. | PK772 | PK_F4 | Mean (±SE) GSK2982772 Plasma Concentration Data by time Relative to Dose by Study Day | Mean concentration vs time (pre-dose =0, 1, 2, 4, and 6 hours post dose) for Day 1, 8 and 43. One plot/panel per regimen (bid and tid) | SAC [1] |
| 4.5. | PK772 | PK_F5 | Mean (±SE) GSK2982772 Plasma Concentration Data by Time relative to Dose, by Dosing Regimen | Mean concentration vs time for bid and tid regimen on one plot. One panel per day (1, 8 and 43) | AR<br>SAC [1] |
| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.6. | PK772 | PK_F1 | GSK2982772 Trough Concentrations in Plasma and Synovial Fluid by Study Day | Spaghetti Plot of observed trough concentrations by body fluid (plasma and synovial fluid) on Day 43 and D85. One panel each for BID and TID Just present subjects who have both plasma and synovia concentrations and update x-axis label to say concentration use legend to distinguish between synovial and plasma concentration | SAC [1] |
| 4.7. | PK772 | PK_F6 | GSK2982772 Trough Concentrations Plasma vs Synovial Fluid | Scatter plot of GSK2982772 Trough Plasma Concentration on X-axis and synovial fluid concentration on Y-Axis. All data, one symbol each for bid and tid Only include subjects who have both plasma and synovial concentration data | AR<br>SAC [1] |

# 12.10.11. Pharmacokinetic/Pharmacodynamic Figures

| PK/PD | PK/PD Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1. | PK772 | PK_F6 | GSK2982772 Plasma Trough Concentration vs Blood TEAR1% Target engagement by Study Day | Scatter plot of GSK2982772 Trough Plasma Concentration vs Blood TEAR1. All data on one plot, one symbol each for bid and tid | SAC [1] |
| 5.2. | PK772 | PK_F6 | GSK2982772 Synovial Fluid Trough Concentration vs Synovial Fluid TEAR1% Target engagement | Scatter plot of GSK2982772 Trough<br>Synovial Fluid Trough Concentration vs<br>Synovial Fluid TEAR1. All data on one<br>plot, one symbol each for bid and tid | SAC [1] |
| 5.3. | PK772 | PK_F6 | GSK2982772 Plasma Trough Concentration vs DAS28 (CRP)<br>Change from baseline | Scatter plot of GSK2982772 Trough Plasma Concentration vs DAS28 change from baseline. All data on one plot, one symbol each for bid and tid, separate page for each relevant visit | SAC [1] |

# 12.10.12. Biomarker Tables

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Inflamn | natory Biomark | ers in blood | | | |
| 6.1. | Safety | PD_T1 | Summary of Blood Inflammatory Biomarkers | One page for each cell type/measure by visit/time and treatment | SAC [1] |
| 6.2. | Safety | PD_T2 | Summary of Percentage Change from Baseline in Blood Inflammatory Biomarkers | One page for each cell type/measure by visit/time and treatment | SAC [1] |
| 6.3. | Safety | PD_T3 | Adjusted Mean (95% CI) Percentage Change in Blood Inflammatory Biomarkers | Present %CVb instead of SE | SAC [1] |
| 6.4. | Safety | PD_T1 | Summary of Blood Inflammatory Biomarkers by Dosing Regimen | One page for each cell type/measure by visit/time and treatment/dosing regimen | SAC [1] |
| 6.5. | Safety | PD_T2 | Summary of Percentage Change from Baseline in Blood Inflammatory Biomarkers by Dosing Regimen | One page for each cell type/measure by visit/time and treatment/dosing regimen | SAC [1] |
| 6.6. | Safety | PD_T3 | Adjusted Mean (95% CI) Percentage Change in Blood Inflammatory Biomarkers by Dosing Regimen | Present %CVb instead of SE<br>Separate page for each dosing regimen | SAC [1] |
| Pathwa | y and Target e | ngagement | | | |
| 6.7. | Safety | EFF_T1 | Summary of TEAR1 % Target Engagement in Blood | | SAC [1] |
| 6.8. | Safety | PD_T4 | Adjusted Mean (95% CI) TEAR1 % Target Engagement in Blood | | SAC [1] |
| 6.9. | Safety | EFF_T1 | Summary of Pathway Engagement in Blood | No longer being produced due to limited sample size | SAC [1] |

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| mRNA | | | | | |
| 6.10. | Safety | PD_T2 | Summary of mRNA Intensity of Inflammatory Gene Transcripts in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. | SAC2 [1] |
| 6.11. | Safety | PD_T5 | Frequency Table Summarising the Number of Probe Sets with Various Fold Change in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. Use cut-offs 1.5 and -1.5 initially. Change to -1.25 and 1.5 if no one achieves the initial cut-offs | SAC2 [1] |
| 6.12. | Safety | PD_T6 | Summary of Analysis for Microaray mRNA Intensity Data in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. If Adj Mean FC lies between -1 and 1 then do not include on table | SAC2 [1] |
| 6.13. | Safety | PD_T2 | Summary of mRNA Percentage Inhibition of Inflammatory<br>Gene Transcripts in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. | SAC2 [1] |
| 6.14. | Safety | PD_T6 | Summary of Analysis for Microaray mRNA Percentage Inhibition Data in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. If Adj Mean FC lies between -1 and 1 then do not include on table | SAC2 [1] |

# 12.10.13. Biomarker Figures

| Pharma | Pharmacodynamic (and or Biomarker): Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1. | Safety | EFF_F1 | Inflammatory Blood Biomarkers, Adjusted Mean (±SE) Change from Baseline in and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | One page for each cell type/measure by visit/time and treatment | SAC [1] |
| 6.2. | Safety | EFF_F2 | Individual Subject Profiles of Inflammatory Biomarkers | Separate page for each cell type/measure | SAC [1] |
| 6.3. | Safety | EFF_F1 | Inflammatory Blood Biomarkers, Adjusted Mean (±SE) Change from Baseline in and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment and Dosing regimen over Time | One page for each cell type/measure by visit/time and treatment/dosing regimen | SAC [1] |
| 6.4. | Safety | EFF_F1 | TEAR1 % Target Engagement in Blood, Adjusted Mean (±SE) Change from Baseline in and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time | | SAC [1] |
| 6.5. | Safety | PD_F1 | Individual Subject Profiles for mRNA Expression of Inflammatory Gene Transcripts in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. Line plot by subjid coloured by treatment group for each probeset / gene. | SAC2 [1] |
| 6.6. | Safety | PD_F2 | Adjusted Mean Intensities for mRNA Expression of Inflammatory Gene Transcripts in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. Y xais – log2 scale | SAC2 [1] |

| Pharma | Pharmacodynamic (and or Biomarker): Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.7. | Safety | PD_F3 | Adjusted Mean (±SE) Fold Change in mRNA Expression of Inflammatory Gene Transcripts in Blood | GSK to produce Only to be produced for significant probsets based on adjusted p-values. If Adj Mean FC lies between -1 and 1 then do not include on table Include band from FC -1 to 1, transparency 0.5 | SAC2 [1] |

# 12.10.14. ICH Listings

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | • | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC[1] |
| 2. | Randomised | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC[1] |
| 3. | Randomised | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC[1] |
| 4. | Randomised | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC[1] |
| Protoc | ol Deviations | | | | |
| 5. | Randomised | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC[1] |
| 6. | Randomised | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC[1] |
| Popula | ations Analysed | | | | |
| 7. | All Subjects | SP3/SP3a | Listing of Subjects Excluded from Any Population | ICH E3 | SAC[1] |
| Demog | graphic and Bas | seline Characteristic | CS | | |
| 8. | Randomised | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC[1] |
| 9. | Randomised | POP_L1 | Listing of Rheumatoid Arthritis Disease History | Include time since formal diagnosis of RA and time since onset of first musculoskeletal symptoms | SAC[1] |
| 10. | Randomised | DM9 | Listing of Race | ICH E3 | SAC[1] |
| 11. | Randomised | MH2 | Listing of Medical History (including CV risk factors) | IDSL | SAC[1] |
| Prior a | nd Concomitan | t Medications | | • | |
| 12. | Randomised | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC[1] |

| ICH: Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | ure and Treatmo | ent Compliance | | | |
| 13. | Randomised | EX3 | Listing of Exposure Data | ICH E3 Please add a column for study treatment to differentiate between dates/times for IP and Methotrexate | SAC[1] |
| 14. | Randomised | POP_L2 | Listing of Dispensing Data | Listing of container number, number of tablets dispensed, returned and then %compliance | SAC[1] |
| Advers | se Events | | | | |
| 15. | Randomised | AE8 | Listing of All Adverse Events | ICH E3 | SAC[1] |
| 16. | Randomised | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC[1] |
| 17. | Randomised | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC[1] |
| Seriou | s and Other Sig | nificant Adverse E | vents | | |
| 18. | Randomised | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | SAC[1] |
| 19. | Randomised | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC[1] |
| 20. | Randomised | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC[1] |
| 21. | Randomised | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC[1] |
| 22. | Randomised | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data:<br>Event and Description (Section 1- Section 2) | IDSL | SAC [1] |
| 23. | Randomised | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | IDSL | SAC [1] |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Randomised | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | IDSL | SAC [1] |
| 25. | Randomised | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5- Section 8) | IDSL | SAC [1] |
| Hepato | biliary (Liver) | | | | |
| 26. | Randomised | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | IDSL | SAC[1] |
| 27. | Randomised | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | IDSL | SAC[1] |
| All Lab | oratory | | | , | |
| 28. | Randomised | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC[1] |
| 29. | Randomised | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC[1] |
| 30. | Randomised | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC[1] |
| 31. | Randomised | UR2A | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC[1] |
| 32. | Randomised | LB5 | Listing of Lipids Outside of the Normal Range | Include fasted status. | IA [1], SAC[1] |
| ECG | | | | · | |
| 33. | Randomised | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL Include absolute PCI subjects. Footnote: H=High absolute, L= Low absolute | SAC[1] |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 34. | Randomised | EG3 | Listing of All ECG Changes for Subjects with a Value of Potential Clinical Importance | Include change from baseline PCI subjects. Footnote: H=High change from baseline value, L= Low change from baseline value | SAC[1] |
| 35. | Randomised | EG3 | Listing of ECG Values of Potential Clinical Importance | "Include absolute PCIs. Footnote: H=High absolute, L= Low absolute." | SAC[1] |
| 36. | Randomised | EG3 | Listing of ECG Changes of Potential Clinical Importance | "Include change from baseline PCIs. Footnote: H=High change, L= Low change." | |
| 37. | Randomised | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL | SAC[1] |
| 38. | Randomised | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC[1] |
| Vital Si | igns | | | | |
| 39. | Randomised | VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC[1] |
| 40. | Randomised | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC[1] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 85 | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC[1] |

# 12.10.15. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CSSRS | <b>;</b> | | | | |
| 41. | Randomised | ECSSRS4 | Listing of C-SSRS suicidal Ideation and Behaviour Data | | SAC[1] |
| 42. | Randomised | ECSSRS5 | Listing of C-SSRS Suicidal Behaviour Details | | SAC[1] |
| PK | | | | | |
| 43. | PK772 | PK07 | Listing of GSK2982772 Pharmacokinetic Concentration-Time Data | | SAC[1] |
| 44. | PKMeth | PK07 | Listing of Methotrexate Pharmacokinetic Concentration-Time Data | | SAC[1] |
| Efficac | ;y | | | | |
| 45. | Randomised | EFF_L11 | Listing of FACIT-Fatigue | | SAC[1] |
| 46. | Randomised | EFF_L8 | Listing of HAQ-DI | | SAC[1] |
| 47. | Randomised | EFF_L10 | Listing of Patient and Physician Global Assessment | | SAC[1] |
| 48. | Randomised | EFF_L6 | Listing of DAS28-CRP, EULAR response and Joint Counts | | SAC[1] |
| 49. | Randomised | EFF_L7 | Listing of ACR Response Rates and ACR Components | | SAC[1] |
| 50. | Randomised | EFF_L1 | Listing of MRI Data, Inflammatory Structural Joint Damage: RAMRIS | | SAC[1] |
| 51. | Randomised | EFF_L2 | Listing of MRI, Inflammatory Structural Joint Damage: RAMRIQ | | SAC[1] |
| 52. | Randomised | EFF_L3 | Listing of MRI, Inflammatory Structural Joint Damage: CARLOS | | SAC[1] |
| 53. | Randomised | EFF_L4 | Listing of Joint Inflammation: DCE-MRI | | SAC[1] |
| 54. | Randomised | EFF_L5 | Listing of Swollen and Tender Joint States | | SAC[1] |
| 55. | Randomised | EFF_L12 | Listing of Patient Assessment of Joint Pain | | SAC[1] |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 56. | Randomised | EFF_L9 | Listing of RA Symptom and Impact Diary | | SAC[1] |
| 57. | Safety | n/a | Raw SAS Output of Statistical Analysis of FACIT-Fatigue | | SAC[1] |
| 58. | Safety | n/a | Raw SAS Output of Statistical Analysis of HAQ-DI | | SAC[1] |
| 59. | Safety | n/a | Raw SAS Output of Statistical Analysis of Patient Global Assessment | | SAC[1] |
| 60. | Safety | n/a | Raw SAS Output of Statistical Analysis of Physician Global Assessment | | SAC[1] |
| 61. | Safety | n/a | Raw SAS Output of Statistical Analysis of DAS28(CRP) | | SAC[1] |
| 62. | Safety | n/a | Raw SAS Output of Statistical Analysis of DAS28(CRP) by dosing regimen | | SAC[1] |
| 63. | Safety | n/a | Raw SAS Output of Statistical Analysis of TJC(28) | | SAC[1] |
| 64. | Safety | n/a | Raw SAS Output of Statistical Analysis of SJC(28) | | SAC[1] |
| 65. | Safety | n/a | Raw SAS Output of Statistical Analysis of MRI:RAMRIS | | SAC[1] |
| 66. | Safety | n/a | Raw SAS Output of Statistical Analysis of MRI:RAMRIQ | | SAC[1] |
| 67. | Safety | n/a | Raw SAS Output of Statistical Analysis of MRI:CARLOS | | SAC[1] |
| 68. | Safety | n/a | Raw SAS Output of Statistical Analysis of DCE-MRI | | SAC[1] |
| 69. | Safety | n/a | Raw SAS Output of Statistical Analysis of DCE-MRI by Dosing Regimen | | SAC[1] |
| 70. | Safety | n/a | Raw SAS Output of Statistical Analysis of Patient Assessment of joint pain | | SAC[1] |
| 71. | Safety | n/a | Raw SAS Output of Statistical Analysis of CRP | | SAC[1] |
| 72. | PP | n/a | Raw SAS Output of Statistical Analysis of DAS28(CRP) | | SAC[1] |

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 73. | PP-completers | n/a | Raw SAS Output of Statistical Analysis of DAS28(CRP)-PP completers | Include subjects that complete the study and are in the PP population | SAC[1] |
| 74. | Safety | n/a | Raw SAS Output of Statistical Analysis of CDAI | | AR, SAC[1] |
| 75. | Safety | n/a | Raw SAS Output of Statistical Analysis of SDAI | | AR, SAC[1] |
| Bioma | rker | | | • | |
| 76. | Randomised | PD_L1 | Listing of Inflammatory Biomarkers in Blood | | SAC[1] |
| 77. | Randomised | PD_L3 | Listing of TEAR1 % Target Engagement in Blood | | SAC[1] |
| 78. | Randomised | PD_L3 | Listing of TEAR1 % Target Engagement in Synovial Tissue | | SAC[1] |
| 79. | Randomised | | Listing of Pathway Engagement in Blood | No longer being produced due to limited sample size | SAC[1] |
| 80. | Randomised | PD_L2 | Listing of mRNA Expression of Inflammatory Gene Transcripts in Blood | Only to be produced for significant probsets based on adjusted p-values. GSK To produce | SAC2[1] |
| 81. | Safety | n/a | Raw SAS Output of Statistical Analysis of Blood Inflammatory Biomarkers | | SAC[1] |
| 82. | Safety | n/a | Raw SAS Output of Statistical Analysis of Blood Inflammatory Biomarkers by Dosing Regimen | | SAC[1] |
| 83. | Safety | n/a | Raw SAS Output of Statistical Analysis of TEAR1 Target Engagement in Blood | | SAC[1] |
| 84. | Safety | n/a | Raw SAS Output of Statistical Analysis of mRNA in Blood | GSK To produce | SAC2[1] |

# 12.11. Appendix 13: Example Mock Shells for Data Displays

Example:
POP\_L1
Pop\_L1

Protocol: 203168

Population: Randomised

Listing of RA Disease History

| Treatment Group | Site ID/ Unique<br>Subject ID | Date of formal diagnosis | Time since formal diagnosis (years) | Date of onset of first musculoskeletal symptoms | Time since onset of first musculoskeletal symptoms (years) |
|---|---|---|---|---|---|
| GSK2982772 | XX/XXXXX | DDMMMYYY | xx.x | DDMMMYYY | xx.x |
| | XX/XXXXX | DDMMMYYY | xx.x | DDMMMYYY | xx.x |
| | XX/XXXXX | DDMMMYYY | xx.x | DDMMMYYY | xx.x |

## 203168

Example:POP\_L2

Page 1 of

n

Protocol: 203168

Population: Randomised

## Listing of Dispensing Data

| Treatment Group | Site ID/ Unique<br>Subject ID | Visit | Container number | Number of<br>tablets<br>dispensed | Number of<br>tablets<br>returned | Treatment<br>Compliance<br>(%) <sup>1</sup> |
|---|---|---|---|---|---|---|
| GSK2928772 | XX/XXXXX | Day 1 | XXXXXX | XX | XX | |
| | | | XXXXXX | XX | XX | |
| | | | XXXXXX | XX | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | Day 29 | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | Day 57 | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |
| | | | XXXXXX | xx | XX | |

| 203168 | | | - | | |
|--------|----|----|--------|-------|----------|
| | xx | xx | XXXXXX | | |
| | XX | XX | XXXXXX | | |
| XX.X | XX | XX | XXXXXX | | |
| | xx | XX | XXXXXX | Day 1 | XX/XXXXX |
| | • | • | • | | |

## PPD

Note: Compliance will only be calculated for subjects who took at least one dose.

<sup>&</sup>lt;sup>1</sup> Compliance = (Total tablets taken/total tablets expected to be taken) \*100.

Example EFF\_T1 

Example EFF\_T1
Protocol: 203168
Population: Safety

Table XX: Summary Statistics for [Continuous Parameter] by Treatment and Visit

| | | | | | {95% CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | N | Visit | n | Mean | (Lower, Upper)} | SD | Median | Min. | Max. |
| Placebo | 18 | Day X | 18 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | xxxx.xx | xxxx.x | XXXX.X |
| | | Day Y | 18 | XXXX.XX | (xxxx.xx,xxxxxxx) | XX.XX | XXXX.XX | XXXX.X | XXXX.X |
| | | Day Z | 18 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| GSK2982772 | 6 | Day X | 6 | xxxx.xx | (xxxx.xx,xxxx) | XX.XXX | xxxx.xx | xxxx.x | XXXX.X |
| | | Day Y | 6 | xxxx.xx | (xxxx,xxxxxx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| | | Day Z | 6 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |

Example EFF\_T2 

Protocol: 203168
Population: Safety

PPD

Table XX: Summary Statistics for Change from Baseline in [Continuous Parameter] by

Treatment and Visit

| | | | | | {95% CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | N | Visit | n | Mean | (Lower, Upper)} | SD | Median | Min. | Max. |
| Placebo | 18 | Day X | 18 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| | | Day Y | 18 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| | | Day Z | 18 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| GSK2982772 | 6 | Day X | 6 | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xxx | XXXX.XX | xxxx.x | xxxx.x |
| | | Day Y | 6 | XXXX.XX | (xxxx,xxxxxxxx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| | | Day Z | 6 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| | | | | | , | | | | |

90

203168

Example: EFF\_T3
Protocol: 203168

Protocol: 203168 Page 1 of x Population: Safety

Table x.x:

Repeated Measures Analysis of the Change from Baseline in [Continuous Parameter]

| Visit | Treatment<br>Group | N | n<br> | LSMean[1] | Standard<br>Error | 95% CI for LSMean (Lower, Upper) | Difference<br>from<br>Placebo | 95% CI for<br>Difference<br>(Lower, Upper) |
|---|---|---|---|---|---|---|---|---|
| Day XX | Placebo<br>GSK2982772 | xx | | x.xx<br>x.xx | x.xxx<br>x.xxx | (x.xx, x.xx)<br>(x.xx, x.xx) | x.xx | (x.xx, x.xx) |
| Day XX | Placebo<br>GSK2982772 | xx | | x.xx<br>x.xx | x.xxx<br>x.xxx | (x.xx, x.xx)<br>(x.xx, x.xx) | x.xx | (x.xx, x.xx) |

. . .

Repeated Measures Analysis adjusted for Baseline Score, Treatment Group, Visit, Baseline Score by Visit and Treatment Group

by Visit Interaction

[1] LSMean is least squares adjusted mean.

Example: EFF\_T4
Protocol: 203168
Population: Safety


## Summary of DAS28(CRP) EULAR Response Categories

| | | Treatment AN=xx | Treatment B<br>N=xx |
|-------|--------------------|-----------------|---------------------|
| Visit | EULAR Category [1] | n % (SE) | n % (SE) |
| Day X | n | XX | xx |
| | No response | Xx xx (xx) | xx xx (xx) |
| | Moderate Response | xx xx (xx) | xx xx (xx) |
| | Good Response | xx xx(xx) | xx xx (xx) |

<sup>[1]</sup> Response at a given time point is defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to baseline.

Example: EFF T5 Protocol: 203168

Population: Safety

Summary of ACR Response Rates [1]

| ACR20 | | | |
|---|---|---|---|
| | | Treatment A | |
| Visit | | N=xx | $\begin{array}{c} \texttt{Treatment B} \\ \texttt{N=} \texttt{xx} \end{array}$ |
| | | n % (SE) | n % (SE) |
| Day X | n | XX | |
| | No Response | xx xx (xx) | XX xx xx (xx) |
| | Response | xx xx (xx) | xx xx (xx) |
| DAY Y | n | xx | xx |
| | No Response | xx xx (xx) | xx xx (xx) |
| | Response | xx xx (xx) | xx xx (xx) |

<sup>[1]</sup> The American College of Rheumatology's (ACR) definition for calculating improvement in RA is calculated as a 20% improvement (ACR20) in both tender and swollen joint counts and 20% improvement in at least 3 of the 5 remaining ACR-core set measures: patient and physician global assessments, patient's assessment of arthritis pain, disability (HAQ-DI), and an acute-phase reactant (i.e. CRP value). Similarly, ACR50 and ACR70 are calculated with the respective percent improvement.

#### PPD

Example: EFF T6 Protocol: 203168


## Population: Safety

Table XX Summary of Bayesian Analysis of Change from Baseline in DAS28-CRP at day 85

| | | | Probabil | lity (trea | tment diffe | erence > x | ), |
|---|---|---|---|---|---|---|---|
| Treatment | SD of Treatment | 95% Credible | | whe | ere x = | | |
| Difference | Difference | Interval [1] | 0 | 0.3 | 0.5 | 0.7 | 1 |
| x.xx | x.xx | ( x.xx, x.xx) | <br>xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |

A non-informative prior for the change in DAS28-CRP score from baseline in each treatment group was used, thus maximising the information provided by the observed data; the prior follows a Normal  $(0,10^36)$  distribution.

Note: A reduction in score on the DAS28-CRP scale is associated with disease improvement. The probability statements above are shown on the positive scale, representing a difference in decline, therefore the larger the difference in decline the greater the improvement over placebo.

[1] Interval is defined as the 2.5th and 97.5th percentiles of the posterior distribution.

203168

Example: EFF\_T7
Protocol: 203168


Population: Safety

Table XX Summary of Bayesian Analysis of ACR20 at day 85

| Treatment | SD of Treatment | 95% Credible | Probak | <b>-</b> · | eatment dif<br>where x = | ference > x | <b>(</b> ), |
|---|---|---|---|---|---|---|---|
| Difference | Difference | Interval [1] | 0 | 5 | 10 | 20 | 30 |
| xx.x | xx.xx | ( xx.xx, xx.xx) | xx | xx.xx | <br>xx.xx | xx.xx | XX.XX |

An non-informative prior for the probability of acheiving ACR 20 in each treatment group was used, thus maximising the information provided by the observed data; the prior follows a Beta(1,1) distribution.

[1] Credible Interval is defined as the 2.5th and 97.5th percentiles of the posterior distribution.

Example: EFF\_F1 

Protocol: 203168
Population: Safety

[Continuous Parameter,] Adjusted Mean (+/-SE) Change from Baseline and Box and Whisker Plot of Unadjusted Change from Baseline by Treatment over Time



PPD

Example: EFF\_F2
Protocol: 203168 Population: Safety

# 





97

Example: EFF\_F3 Protocol: 203168 Population: Safety


Proportion of subjects in each DAS28-CRP EULAR Response Category




Example: EFF\_F4 Protocol: 203168 Population: Safety

# Proportion of subjects achieving ACR20/50/70



Example: PD\_T1
Protocol: 203167

 Population: Safety

Table X.X

Summary Statistics of Blood Inflammatory Biomarkers

Parameter: X (Units)

| Treatment | N Visit | Planned<br>Relative<br>Time | n | Mean | {95% CI (Lower, Upper)} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Placebo | XX DAY 1 | PRE-DOSE | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | х.х | XX.X |
| | DAY 43 | PRE-DOSE | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | Х.Х | XX.X |
| | DAY 85 | DAY 85 | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | Х.Х | XX.X |
| GSK2982772 | XX DAY 1 | PRE-DOSE | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | Х.Х | XX.X |
| | DAY 43 | PRE-DOSE | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | Х.Х | XX.X |
| | DAY 85 | DAY 85 | XX | X.XX | ( X.XX, X.XX) | X.XXX | X.XX | Х.Х | XX.X |

203168

Example: PD\_T2
Protocol: 203168

Protocol:  $2\overline{0}$ 3168 

Population: Safety

Table X.X

Summary of Percentage Change in Blood Inflammatory Biomarkers

Parameter: X (Units)

| Treatment | N | Vis | it | Mean<br>Baseline<br>[1] | Planned<br>Relative<br>Time | n | Mean | {95% CI (Lower, Upper)} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | XX | DAY | 43 | X.XXX | PRE-DOSE | XX | XX.XXX | ( XX.XXX,XX.XXX) | XXX.XXXX | x.xxx | XX.XX | XX.XX |
| | | DAY | 85 | X.XXX | DAY 85 | XX | XX.XXX | ( XX.XXX,XX.XXX) | XXX.XXXX | X.XXX | XX.XX | XX.XX |
| GSK2982772 | 2 XX | DAY | 43 | X.XXX | PRE-DOSE | XX | XX.XXX | ( XX.XXX,XX.XXX) | XXX.XXXX | X.XXX | XX.XX | XX.XX |
| | | DAY | 85 | X.XXX | DAY 85 | XX | XX.XXX | ( XX.XXX,XX.XXX) | XXX.XXXX | X.XXX | XX.XX | XX.XX |

<sup>[1]</sup> Baseline is taken as the mean of the planned pre-dose measurements.

203168


Example: PD\_T3
Protocol: 203163

Population: Safety

Table X.X

Adjusted Mean (95% CI) Percentage Change in Blood Inflammatory Biomarkers

Parameter: X (Units)

| Visit | N | Treatment | n | Geometric<br>LSMean | e<br>%CVb | 95% CI for<br>LSMean | Difference<br>From<br>Placebo | 95% CI for Difference Lower, Upper) |
|---|---|---|---|---|---|---|---|---|
| DAY 43 | XX | Placebo | XX | XX.XX | XX.XXX | (XX.XX, XX.XX | • | |
| | XX | GSK2982772 | XX | XX.XX | XX.XXX | (XX.XX, XX.XX | ) XX.XX | (XX.XX, XX.XX) |
| DAY 85 | XX<br>XX | Placebo<br>GSK2982772 | XX<br>XX | XX.XX<br>XX.XX | XX.XXX<br>XX.XXX | (XX.XX, XX.XX<br>(XX.XX, XX.XX | • | (XX.XX, XX.XX) |

Note: Baseline is defined as the latest pre-dose assessment.

Note: Analysis performed using a MMRM model, adjusting for the following covariates: treatment, baseline,

Visit, baseline by visit and an interaction between treatment and visit.

203168

Example: PD\_T4


Population: Safety

Table x.x:
Adjusted Mean (95% CI) TEAR1 % Target Engagement in Blood

| | | | SMean_<br>ement | | oo LSMean_<br>agement | Treatment Ratio | Diff % Engagement |
|---|---|---|---|---|---|---|---|
| Visit | Comparison | Ratio | 용 | Ratio | -<br>% | (95% CI) | (95% CI) |
| DAY 43 | GSK2982772<br>vs Placebo | X.XX | Х | X.XX | X | X.XX (X.XX, X.XX) | X.X (X.X, X.X) |
| DAY 85 | GSK2982772<br>vs Placebo | X.XX | Χ | X.XX | X | x.xx (x.xx, x.xx) | X.X (X.X, X.X) |

Note: Baseline is defined as the latest pre-dose assessment.

Note: Percentage target engagement = (1 - engagement ratio) \* 100.

Repeated Measures Analysis adjusted for log baseline, Treatment Group, Visit, log baseline by Visit and

Treatment Group by Visit Interaction

203168


Example: PD\_T5
Protocol: 203168

Population: Safety

Table XX.XX:

Frequency table summarising the number of probe sets in various fold change

| | | | | | | Fold Change | in Blood |
|---|---|---|---|---|---|---|---|
| Probeset | Gene | Visit | N | n | Treatment | < 1.5 | >1.5 |
| XXXXXX | XXXXXX | Baseline | XX | XX | Placebo<br>GSKXXXXXX XXmg | xx (xx.xx)<br>xx (xx.xx) | xx (xx.xx)<br>xx (xx.xx) |
| | | WEEK xx | XX | XX | Placebo<br>GSKXXXXXX XXmg | xx (xx.xx)<br>xx (xx.xx) | xx (xx.xx)<br>xx (xx.xx) |
| | | WEEK xx | XX | XX | Placebo<br>GSKXXXXXX XXmg | xx (xx.xx)<br>xx (xx.xx) | xx (xx.xx)<br>xx (xx.xx) |

Example: PD\_T6
Protocol: 203168


Table XX.XX:
Summary of Analysis for Microarray mRNA Data from xxxx

| | | | | | | Adjusted | 1 | | Fold | Adjusted |
|---|---|---|---|---|---|---|---|---|---|---|
| Probeset | Gene | Visit | N | n | Treatment | mean | 95% | CI | Change | p-value |
| XXXXXX | XXXXXX | Baseline | XX | XX | Placebo | XX.X | (XX.X, | XX.X) | | |
| | | | | | GSKXXXXXX XXmg | XX.X | (XX.X, | XX.X) | XX.X | X.XXX |
| | | WEEK xx | XX | XX | Placebo | xx.x | (XX.X, | XX.X) | | |
| | | | | | GSKXXXXXX XXmg | xx.x | (XX.X, | XX.X) | XX.X | x.xxx |
| | | WEEK xx | XX | XX | Placebo | XX.X | (XX.X, | XX.X) | | |
| | | | | | GSKXXXXXX XXmg | XX.X | (XX.X, | XX.X) | XX.X | X.XXX |

Note: Fold change in relative to the baseline value

Note: Fold change from baseline is defined as ratio to baseline if the ratio is  $\geq 1$ , otherwise it is defined as -1/rratio to baseline.

Programming note: Please present SE not 95% CI

Example: PD\_F1  Protocol: 203168

Protocol: 203168
Population: Safety

Figure X
Individual [Continuous Parameter] Scores over Time by Treatment



Example: PD\_F2

Protocol: 203168 Page 1 of x Population: Safety

Figure XX.XX:
Adjusted mean probe set intensity values (+/- SE) by time from xxxx

## Gene ID: XXXX



Example: PD F3 Protocol: 203168


Population: Safety

# Figure XX.XX: Adjusted Fold Change in mRNA Expression

## Gene ID: XXXX



Programming note to present SE's not 95% CI

Example: EFF\_L1
Protocol: 203168
Population: Safety

Listing of MRI Data, Inflammatory Structural Joint Damage: RAMRIS

Treatment Group: Treatment A

| Site ID/<br>Unique | | Number of<br>Available | | Bone Erosion | Bone Edema/Osteitis | |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Joints | Synovitis | | | Cartilage Loss |
| XXXX/ XXXXX | Baseline | xx | xxx | XXX | Xxx | XXX |
| | Week X<br>Etc. | XX | XXX | XXX | Xxx | xxx |
| xxxx/ xxxxx | Baseline | xx | xxx | XXX | Xxx | xxx |
| | Week X<br>Etc. | XX | XXX | xxx | Xxx | xxx |

203168

Example: EFF\_L2 Page 1 of n Protocol: 203168

Protocol: 203168
Population: Safety

Listing xx

Listing of MRI Data, Inflammatory Structural Joint Damage: RAMRIQ

| Site ID/<br>Unique<br>Subject ID | Visit | Synovitis | Synovitis<br>Normalized | Erosive Damage<br>(Normalized) | Cartilage Space Loss | Bone Marrow<br>Lesions |
|---|---|---|---|---|---|---|
| XXXX/ XXXXX | Baseline<br>Week X<br>Etc. | | | | | |
| XXXX/ XXXXX | Baseline<br>Week X<br>Etc. | | | | | |

DDF

203168


Example: EFF\_L3
Protocol: 203168
Population: Safety

Listing xx

Listing of MRI Data, Inflammatory Structural Joint Damage: CARLOS

Treatment Group: Treatment A

| Site ID/<br>Unique<br>Subject ID | Visit | Result |
|---|---|---|
| XXXX/ XXXXX | Baseline<br>Week X<br>Etc. | Complete cartilage denuding or diffuse bone-on-bone contact<br>Complete ankylosis |
| XXXX/ XXXXX | Baseline<br>Week X<br>Etc. | |


Example: EFF\_L4
Protocol: 203168
Population: Safety

Listing of Joint Inflammation: DCE-MRI

| | | Treatment G | roup: Treatme | ent A | | | |
|---|---|---|---|---|---|---|---|
| | Exchan<br>ge | Interstitial | Plasma<br>Volume | Joint<br>Volume | Enhancing<br>Volumne | Initial Rate | Maximum signal intensity |
| Visit | Rate | Volume | | | | of Enhancement | enhancement |
| Baseli<br>ne<br>Week X<br>Etc. | | | | | | | |
| Baseli<br>ne<br>Week X | | | | | | | |
| | Baseli<br>ne<br>Week X<br>Etc.<br>Baseli<br>ne | ge Visit Rate Baseli ne Week X Etc. Baseli ne Week X | Exchan ge Interstitial Visit Rate Volume Baseli ne Week X Etc. Baseli ne Week X | Exchan ge Interstitial Volume Visit Rate Volume Baseli ne Week X Etc. Baseli ne Week X | ge Interstitial Volume Volume Visit Rate Volume Baseli ne Week X Etc. Baseli ne Week X | Exchan plasma Joint Enhancing Volume Volume Volume Visit Rate Volume Baseli ne Week X Etc. Baseli ne Week X | Exchan ge Interstitial Volume Volume Volume Volume Initial Rate of Enhancement Baseli ne Week X Etc. Baseli ne Week X |

Example: EFF\_L5 Page 1 of n Protocol: 203168

Protocol: 203168
Population: Safety

Listing of Observed Swollen and Tender Joint States

Treatment Group: Treatment A

Site ID/Unique Subject ID: <Site ID/Subject ID>

| Visit | | Joints of Left<br>Extremities | Joints of Right<br>Extremities |
|---|---|---|---|
| Baseline | Tender | Shoulder, Wrist,<br>MCP3, PIP5 | Elbow, PIP5<br>Sternoclavicular,<br>Hip, DIP3 |
| | Swollen<br>Not available | | • , |
| Week X<br>Etc. | | | |
| Baseline<br>Week X<br>Etc. | | | |


Protocol: 203168
Population: Safety

Listing of DAS28-CRP, EULAR response and Joint Counts

Treatment Group: Treatment A

| Site ID/<br>Unique Subject<br>ID | | Remission? | Low disease<br>Activity? | TJC28/ TJC68 | SJC28/ SJC66 |
|---|---|---|---|---|---|
| | Visit | | | | |
| XXXX/ XXXXX | - | Yes | | xx.x/ xx.xx | xx.x/ xx.xx |
| | Baseline | | | xx.x/ xx.xx | xx.x/ xx.xx |
| | Week X | | | Etc. | Etc. |
| | Etc. | | | | |
| XXXX/ XXXXX | | No | | xx.x/ xx.xx | xx.x/ xx.xx |
| | Baseline | | | xx.x/ xx.xx | xx.x/ xx.xx |
| | Week X | | | Etc. | Etc. |
| | Etc. | | | | |

Note: DAS28(CRP) remission is achieved by a DAS28(CRP) value lower than 2.6 and DAS28(CRP) Low Disease Activity is defined as a DAS28 score of  $\leq$  3.2.


Protocol: 203168
Population: Safety

Listing of ACR Response Rates and ACR Components

Treatment Group: Treatment A

| Site ID/ Unique<br>Subject ID | e<br>Visit | TJC68 | SJC66 | PtGA | PhGA | Pt Pain | CRP Value | HAQ-DI | ACR<br>20/50/70<br>Response |
|---|---|---|---|---|---|---|---|---|---|
| , | | | | | | | | | |
| XXXX/ XXXXX | Week 1 | Xx | XX | XX | XX | XX | XX | XX | ACR 50 |
| | Week 2 | Xx | XX | XX | XX | Xx | XX | XX | |
| | Etc. | Xx | XX | XX | XX | Xx | XX | XX | ACR 20 |
| | | | | | | Xx | | | |
| XXXX/ XXXXX | Week 1 | XX | XX | XX | XX | Xx | XX | XX | |
| | Week 2 | Xx | XX | XX | XX | Xx | XX | XX | |
| | Etc. | | | | | | | | |

Note: Listing shows percentage change from Baseline. For all components, negative values represent improvement. Note: ACR20 is achieved for a 20% improvement in both TJC68 and SJC66 and 20% improvement in 3 of the 5 remaining components. ACR50 and ACR70 are defined accordingly.

203168

Page

Example: EFF L8

1 of n

Protocol: 203168
Population: Safety

Listing of HAQ-DI

Treatment Group: Treatment A

Site ID/Unique Subject ID: <Site ID/Subject ID>

| | Dress & | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Groom | Rising | Eating<br>Cut | Walking | Hygiene | Reach | Grip | Activity. | | | HAQ-DI |
| | | | meat/ | | Wash | | Open | | | | SCore |
| | | | Lift | | Body/ | | Car/ | | | Help | |
| | Dress/ | Stand | Cup/ | Walk/ | Have | _ , , | Open | Shop/ | | from | |
| | Wash | up/ Get | Open | Climb | Bath/ | Reach/ | Jar/ | Car/ | Aids or | another | |
| Visit | hair | in Bed | Milk | stairs | Toilet | Bend | Turn Tap | Chores | Equipment | Person | |
| Baseline | 1/3 | 0/2 | 0/2/2 | 1/3 | 0/2/2 | 2/2 | 0/2/1 | 0/2/2 | Crutches | Eating, | XX |
| | | | | | | | | | | Rising | |
| Week X | x/x | x/x | x/x/x | x/x | x/x/x | x/x | x/x/x | x/x/x | XXXXX | XXXXX, | |
| | | | | | | | | | | XXXXX | |
| Etc. | ••• | ••• | | | | | | | | ••• | |

Note: 0 = Without any difficulty. 1 = With some difficulty. 2 = With much difficulty. 3 = Unable to do.

Note: HAQ-DI Pain Sore can be found in Listing 20.

Note: Functional areas in order of the columns are: Dress & Groom, Rising, Eating, Walking, Hygiene, Reach, Grip,

Activity

203168


Example: EFF\_L9
Protocol: 203168
Population: Safety

Listing of RA Symptom and Impact Diary [1]

Treatment Group: Treatment A

| Site ID/<br>Unique<br>Subject<br>ID | Visit | Joint Pain<br>Sitting/<br>Lying/<br>Moving | Joint Pain<br>Walking/<br>Standing/<br>Lifting | Joint<br>Paint<br>at its<br>Worst | Energy/<br>Tired | Stiffness/<br>Morning<br>Stiffness | Morning<br>Stiffness<br>Duration | Joint<br>Stiffness<br>Severity | Had<br>to<br>Rest | Sleep<br>Quality/<br>Affection |
|---|---|---|---|---|---|---|---|---|---|---|
| xx/xxxxx | Day X | 2/5/5 | 4/3/4 | 3 | No<br>Energy/<br>A little<br>of the<br>time | All of the time/ Mild | Less than<br>30 Minutes | Mild | All<br>of<br>the<br>time | Bad/ A<br>little |
| XX/XXXXX | Day Y | 0/4/10 | 2/ 5/ 5 | 10 | Some<br>Energy/<br>All of<br>the time | None of the time/ Very severe | No morning stiffness | Severe | Most<br>of<br>the<br>time | Very<br>Good/<br>Somewhat |
| XX/XXXXX | Day Z | | | | | | 2-4 Hours | | | |
| XX/XXXXX | | | | | | | | | | |

<sup>[1]</sup> Symptoms rated relative to the last 24 hours


Protocol: 203168
Population: Safety

Listing of Patient and Physician Global Assessment [1]

Treatment Group: Treatment A

| Site ID/<br>Unique<br>Subject<br>ID | Visit | Actual Date Study Day | Physician<br>Assessment [1] | Patient<br>Assessment<br>[2] |
|---|---|---|---|---|
| XX/XXXXX<br>XX/XXXXX<br>XX/XXXXX | Day X<br>Day Y<br>Day Z | | XX | XX |
| XX/XXXXX | | | | |

- [1] Physician assessment of disease activity using the visual analogue scale with anchor's "0" (none) to "10" (extremely active).
- [2] Patients assessment of how they feel today, using the visual analogue scale with anchor's "0" (Very good)" to "10" (very poor).

203168


Protocol: 203168
Population: Safety

Listing of Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale [1]

Treatment Group: Treatment A

Site ID/ Unique Subject

| Unique<br>Subject<br>ID | Visit | Actual Date | Study Day | Category | Response | Total<br>Score |
|---|---|---|---|---|---|---|
| XX/XXXXX | Day X | | | I feel fatigued I feel weak all over I feel listless ("washed out") I feel tired I have trouble starting things because I | Not at all A little bit Somewhat Quite a bit Very much | XX |
| | | | | am tired I have trouble finishing things because I am tired I have energy I am able to do my usual activities I need to sleep during the day I am too tired to eat I need help doing my usual activities I am frustrated by being too tired to do the things I want to do I have to limit my social activity because I am tired | A little bit Somewhat Not at all A little bit A little bit Somewhat Quite a bit Not at all Somewhat | |

XX/XXXXX

XX/XXXXX Day Z

XX/XXXXX

[1] A global assessment of disease activity using the a visual analogue scale with anchor's "0" (none) to "10" (extremely active).

| PPD Example: Protocol: Populatio | $20\overline{3}168$ | | | | Page 1 of n |
|---|---|---|---|---|---|
| - | _ | | Listing of Patient Assessment of Joint B | ain [1] | |
| Treatment | Group: Treat | ment A | | | |
| Site ID/<br>Unique<br>Subject | | | | Patient | |
| ID | Visit | Actual Date | Study Day | Assessment | |
| XX/XXXXX<br>XX/XXXXX<br>XX/XXXXX | Day X<br>Day Y<br>Day Z | | | XX | |
| XX/XXXXX | | | | | |

[1] RA pain on average over the past 24 hours: using a visual analogue scale with anchor's "0" (no pain) to "10" (most severe pain).

203168

Example : PD\_L1 Page 1 of n

Protocol : 203168
Population : Safety

Listing XX:
Listing of Raw, Change from baseline and Percent Change in [variable]

| Treatment | Subject | Visit | Visit<br>date | Study<br>day | Histopatholgical<br>Scoring | Raw | Change | Percent<br>Change |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxx | xxx | XX/XX/XX | Day 1 | K16<br>CD3/CD11c<br>CD161<br>Elactase +ve cels<br>epidermal thickness | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | | |
| | | XXX | XX/XX/XX | Day 43 | K16<br>CD3/CD11c<br>CD161<br>Elactase +ve cels<br>epidermal thickness | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X |

203168

Example : PD\_L2 Page 1 of n

Protocol : 203168
Population : Safety

Listing XX:

Listing of Absolute, Percentage Inhibition and Maximum Percentage Inhibition in mRNA Expression

| Gene | Treatment | Subject | Visit | CT1/CT2/<br>CTAVG/<br>Copy<br>Number | Value | Percentage<br>Inhibition<br>[1] | Maximum<br>Percentage<br>Inhibition<br>[2] |
|---|---|---|---|---|---|---|---|
| XXXXGENE | GSKXXXXXX XXmg | XXXX | Screening | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | | |
| | | | Baseline | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |
| | | | Week X | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |

203168

Example PD\_L3
Protocol: 203168

Protocol: 203168
Population: All Subjects
Page 1 of 64

Listing 79

Listing of TEAR1 Concentrations and % Target Engagement: Part B

Treatment: Treatment A

| | | Actual | ************************************** | Planned<br>Relative | | | D-1-1-11 | % Target<br>Engagement |
|---|---|---|---|---|---|---|---|---|
| Subj. | Date | Time | Visit | Time | | (pg/mL) | Ratio[]] | [2] |
| PPD | PPD | 9:42 | DAY 1 | PRE-DOSE | Free | 9.31504 | 0.4670 | |
| | | | | | Total | 19.94849 | | |
| | | 11:51 | DAY 1 | 1.5 HR | Free | 5.11583 | 0.3894 | 16.605 |
| | | | | | Total | 13.13721 | | |
| | | 18:20 | DAY 1 | 8 HR | Free | 8.01224 | 0.3926 | 15.929 |
| | | | | | Total | 20.40949 | | |
| | | 10:09 | DAY 1 | 24 HR | Free | 7.82238 | 0.3761 | 19.456 |
| | | | | | Total | 20.79845 | | |
| | | 9:11 | DAY 14 | PRE-DOSE | Free | 8.06836 | 0.3705 | 20.666 |
| | | | | | Total | 21.77966 | | |
| | | 10:50 | DAY 14 | 1.5 HR | Free | 8.44182 | 0.4155 | 11.012 |
| | | | | | Total | 20.31552 | | |
| | | 17:21 | DAY XX | 8 HR | Free | 7.80388 | 0.3734 | 20.033 |
| | | | | | Total | 20.89901 | | |

Note: Only Tru Culture results are included.

<sup>[1]</sup> Ratio=Free/Total

<sup>[2] %</sup>Target Engagement = 100 - ((ratio post/ ratio pre-dose)\* 100).

Example: PK\_F1

Protocol: 203168
Population: PK772

Page 1 f x

Figure XX.XX: GSK2982772 Trough Plasma Concentration by Study Day



USE THIS SHELL FOR FIG. 4.6 AS WELL.

Example: PK F2

Protocol: 203168
Population: PK772


Figure XX.XX: GSK2982772 Trough Plasma Concentration by Study Day



Example: PK\_F3

Protocol: 203168

Population: PK772






Include Day1, 8 and 43 as separate pages

Example: PK\_F4


Population: PK772

Figure XX.XX: Mean GSK2982772 Plasma Concentration Data by Time Relative to Dose by Study Day



Example: PK F5


Population: PK772

Figure XX.XX: Mean GSK2982772 Plasma Concentration Data by Time Relative to Dose by Randomized Regimen



Example: PK F6

Protocol: 203168 Page 1 of x Population: PK772

Figure XX.XX: GSK2982772 Plasma Trough Concentration vs Blood TEAR1% Target engagement

